## Official Title of Study:

An Open-Label, Single-arm, Multi-Center, Phase 3 Study to Evaluate the Efficacy and Safety of BMS-986165 in Japanese Subjects with Moderate-to-Severe Psoriasis

NCT Number: NCT03924427

Document Date (Date in which document was last revised): May 7, 2020

Page: 1

Protocol Number: IM011066 IND Number: 131,993 EX-US Non-IND EUDRACT N/A

Number:

Date, Version: 07-May-2020, Final Approved v5.0

## Clinical Protocol IM011066

An Open-Label, Single-arm, Multi-Center, Phase 3 Study to Evaluate the Efficacy and Safety of BMS-986165 in Japanese Subjects with Moderate-to-Severe Psoriasis

Short Title: Efficacy and Safety of BMS-986165 in Subjects with Moderate-to-Severe Psoriasis

#### **Revised Protocol 04**

Based on the Protocol IM011066, version 4.0, dated 11-Feb-2019 Amendment



**24-hr Emergency Telephone Number** 

North America:

Asia-Pacific:

Bristol-Myers Squibb Research and Development

3401 Princeton Pike Lawrenceville, NJ 08648 6-5-1 Nishi-Shinjuku, Shinjuku-ku, Tokyo, 163-1328, Japan

This document is the confidential and proprietary information of Bristol-Myers Squibb Company and its global affiliates (BMS). By reviewing this document, you agree to keep it confidential and to use and disclose it solely for the purpose of assessing whether your organization will participate in and/or the performance of the proposed BMS sponsored study. Any permitted disclosures will be made only on a confidential "need to know" basis within your organization or to your independent ethics committee(s). Any other use, copying, disclosure or dissemination of this information is strictly prohibited unless expressly authorized in writing by BMS. Any supplemental information (eg, amendments) that may be added to this document is also confidential and proprietary to BMS and must be kept in confidence in the same manner as the contents of this document. Any person who receives this document without due authorization from BMS is requested to

return it to BMS or promptly destroy it. All other rights reserved. References to BMS in this protocol may apply to partners to which BMS has transferred obligations, eg, a Contract Research Organization.

# **DOCUMENT HISTORY**

| Document | Date of Issue | Approver(s) | Summary of Change |
|---|---|---|---|
| Original Protocol | 27-June-2018 | | Not applicable |
| Amendment 01 | 16-Nov-2018 | | <ul> <li>Further clarified the diagnoses parameters for subjects with PsA, GPP, and EP.</li> <li>Updated contact information</li> <li>Corrected minor procedural and typographic errors.</li> <li>Updated Appendix 3 to be consistent with all BMS-986165 studies</li> </ul> |
| Amendment 02 | 08-Jan-2019 | | <ul> <li>Revised certain exclusion criteria (eg, criteria related to urine drug screen and thyroid-stimulating hormone) to be consistent with the global Phase 3 study, BMS-986165 IM011046</li> <li>Corrected minor procedural and typographic errors.</li> </ul> |
| Amendment 03 | 11-Feb-2019 | | Aligned the HBV testing and the related exclusion criterion to the most recent guidelines for the Management of HBV Infection provided by the Japan Society of Hepatology |

| Revised Protocol 04 | 07-May-2020 | Made the following updates: |
|---|---|---|
| (im011066-<br>revprot04) | | Added infection,<br>cardiovascular and<br>suicidal ideation and<br>behavior (SIB)<br>adjudication<br>committees to the study |
| | | Provided clarifications in the protocol to aid sites and subjects in the conduct of the study |
| | | Corrected typographical errors |

#### **SUMMARY OF CHANGES**

#### **Rationale:**

The primary purpose of this global revised protocol is to add the infection, cardiovascular, and suicidal ideation and behavior adjudication committees to the study to align with other studies in the psoriasis program.

Key modifications and clarifications are summarized as follows:

o Added clarifying detail to several items in the protocol

0

Substantive changes made to the previous version of the global protocol and the rationale for these changes are noted below in the summary of key changes table. All changes applied to the protocol body were applied to the synopsis, as necessary; synopsis changes are not included in the summary of key changes table. Only major additions and deletions are provided in this summary document; all minor grammatical, formatting, stylistic changes, or clarifications as well as organizational changes are not included.

| <b>Protocol Section</b> | Revised Protocol Text | Rationale for Change |
|---|---|---|
| 4.1.6.1 Infection<br>Adjudication<br>Committee | Addition of the following Adjudication Committees: An independent Infection Adjudication Committee, composed of individuals with relevant expertise, will blindly review and adjudicate infection AEs, such as opportunistic infections, influenza, herpes zoster, and TB, reported in the study per criteria specified in a separate charter. Additional information about these infections may be collected on the case report form (CRF) in order to characterize and understand them. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee members will not be investigators on the study. | |
| 4.1.6.2<br>Cardiovascular<br>Adjudication<br>Committee | An independent cardiovascular (CV) Adjudication Committee, composed of individuals with relevant expertise, will blindly review and adjudicate cardiovascular and cerebrovascular AEs such as, but not limited to, Major Adverse Cardiovascular Events (MACE) that include death, non-fatal myocardial infarction, non-fatal stroke; revascularization procedures; heart failure; dysrhythmias; heart blocks; and thrombotic events reported in the study per criteria specified in a separate charter. Additional information about cardiovascular and cerebrovascular AEs may be collected on the CRF in order to characterize and understand them. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee members will not be investigators on the study. | Addition of 3 adjudication committees to align with other Phase 3 studies in the psoriasis program which include these committees |
| 4.1.6.3 Suicidal<br>Ideation and<br>Behavior (SIB)<br>Adjudication<br>Committee | An independent Suicidal Ideation and Behavior Adjudication Committee, composed of individuals with relevant expertise, will blindly review and adjudicate suicidal ideation/behavior reported in the study per criteria specified in a separate charter. Additional information about suicidal ideation/behavior may be collected on the CRF. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee members will not be investigators on the study. | |
| 5.3 Lifestyle<br>Restrictions | Updated text: General skin care measures (with above restrictions for topical treatments) that are standard for subjects with plaque psoriasis are permitted. | To clarify general skin care measures used in the trial |

| <b>Protocol Section</b> | Revised Protocol Text | Rationale for Change |
|---|---|---|
| | Updated or added text: 6) Any use of oral psoriasis medications (eg, methotrexate, cyclosporine, retinoids, fumaric acid derivatives) for any indication | |
| | <ul> <li>a. For subjects with generalized pustular psoriasis, one of<br/>the following agents is permitted: cyclosporine, methotrexate,<br/>or retinoids.</li> </ul> | |
| | b. For subjects with erythrodermic psoriasis, concomitant use of cyclosporine is permitted until Week 2. | |
| | 7) Any use of oral <b>or injectable</b> corticosteroids (eg, prednisone, methylprednisolone), unless it is considered necessary for the subject's welfare and/or treatment of an AE/SAE | |
| | <ul> <li>a. For subjects with erythrodermic psoriasis or generalized pustular psoriasis, use of prednisone or its equivalent at a daily dose ≤ 10 mg/day is permitted.</li> </ul> | |
| 6.7.1 Prohibited and/or Restricted | b. Otic, ophthalmic, nasal, or inhaled corticosteroids within recommended doses and with no systemic effects are permitted. | |
| Treatments | 8) Any topical medications/treatments, which are used for any indication, that could affect psoriasis evaluation (including, but not limited to, ultra-high to moderate potency corticosteroids (WHO Classes I-V), >3% salicylic acid, urea, alpha- or beta-hydroxyl acids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, picrolimus, and tacrolimus). | Added clarifying detail around these prohibited medications |
| | Exception: The following topical treatments may be initiated only at Week 24 per investigator's discretion in subjects who have (See Section 4.1.4): | |
| | Ultra-high to moderate potency corticosteroids (Classes I-V), >3% salicylic acid, urea, alpha- or beta-hydroxyl acids, anthralin, calcipotriene, vitamin D derivatives, retinoids, tazarotene | |
| | Note: Low potency topical steroids (WHO Classes VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha- or beta hydroxy acids or other ingredients which are pharmacologically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit. | |
| 6.7.2 Permitted<br>Concomitant<br>Medications | Low potency topical steroids (WHO Classes VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha- or beta-hydroxy acids or other ingredients which are pharmacologically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit. | Added clarifying detail around these medications |

| Protocol Section | Revised Protocol Text | Rationale for Change |
|---|---|---|
| 8.4.5 Clinical<br>Safety Laboratory<br>Assessments | Added the following tests under the Other Analyses section: Serum Immunoglobulin Levels (IgM, IgG, IgA, IgE) | Addition of tests to harmonize with all other Phase 3 studies in the psoriasis program |
| 8.4.7 Suicidal<br>Ideation and<br>Behavior<br>Monitoring | Subjects who answer yes to Questions 4 or 5 which indicates a suicidal ideation severity level of 4 or 5 or document suicidal behavior or suicidal attempts on the eC-SSRS will have their treatments discontinued and be immediately referred to a mental health professional for further evaluation. | Clarified to sites to what levels of suicidal ideation Questions 4 and 5 refer |
| 9.5.1 Adverse<br>Events | Treatment-emergent adverse events (TEAEs), SAEs and deaths, AEs leading to study treatment discontinuation, AEs by maximum severity, and AEs by relationship will be summarized by the MedDRA system organ class and preferred term. All TEAEs as well as each AE-adjudicated category (ie, infections, cardiovascular, and SIB) will also be summarized by preferred term sorted by decreasing frequency. | Added the summarization of these categories because of the addition of the adjudication committees |

# **TABLE OF CONTENTS**

| | PAGE | |
|---|---|---|
| <b>DOCUN</b> | MENT HISTORY | 3 |
| SUMM | ARY OF CHANGES | 5 |
| <b>TABLE</b> | OF CONTENTS | |
| 1 | PROTOCOL SUMMARY | 12 |
| 1.1 | Synopsis | 12 |
| 1.2 | Schedule of Activities (SOA) | 15 |
| 2 | INTRODUCTION | 31 |
| 2.1 | Study Rationale | 31 |
| 2.2 | Background | 32 |
| 3 | OBJECTIVES AND ENDPOINTS | 34 |
| 4 | STUDY DESIGN | 37 |
| 4.1 | Overall Design | 37 |
| 4.2 | Number of Subjects | |
| 4.3 | End of Study Definition | |
| 4.4 | Scientific Rationale for Study Design | |
| 5 | STUDY POPULATION | 41 |
| 5.1 | Inclusion Criteria | 41 |
| 5.2 | Exclusion Criteria | 42 |
| 5.3 | Lifestyle Restrictions | 48 |
| 5.4 | Screen Failures | 48 |
| 6 | TREATMENT | 49 |
| 6.1 | Treatments Administered | 49 |
| 6.2 | Method of Treatment Assignment | 50 |
| 6.3 | Blinding | 50 |
| 6.4 | Dosage Modification | 50 |
| 6.5 | Preparation/Handling/Storage/Accountability | 50 |
| 6.6 | Treatment Compliance | |
| 6.7 | Concomitant Therapy | 51 |
| 6.8 | Treatment After the End of the Study | 53 |
| 7 | DISCONTINUATION CRITERIA | 53 |
| 7.1 | Discontinuation from Study Treatment | 53 |
| 7.2 | Discontinuation from the Study | 55 |
| 7.3 | Lost to Follow-up | |
| 8 | STUDY ASSESSMENTS AND PROCEDURES | 56 |
| 8.1 | Efficacy Assessments | 56 |
| 8.2 | Adverse Events | |
| 8.3 | Overdose | 65 |
| 8.4 | Safety | <u>65</u> |
| 8.8 | Health Economics OR Medical Resource Utilization and Health Economics | 73 |

| 9 | STATISTICAL CONSIDERATIONS | 73 |
|---|---|---|
| 9.2 | Populations for Analyses | 73 |
| 9.3 | Endpoints | 73 |
| 9.4 | Efficacy Analyses | |
| 9.5 | Safety Analyses | |
| 9.6 | Other Analyses | |
| 9.7 | Interim Analysis | 77 |
| 10 | REFERENCES | |
| 11 | APPENDICES | 82 |
| APPENDE | IX 1 ABBREVIATIONS AND TRADEMARK | XS83 |
| APPENDE | IX 2 STUDY GOVERNANCE CONSIDERAT | ΓΙΟΝS88 |
| APPENDE | IX 3 ADVERSE EVENTS AND SERIOUS AI | OVERSE EVENTS: |
| | <b>DEFINITIONS AND PROCEDURES FO</b> | OR RECORDING, |
| | EVALUATING, FOLLOW-UP AND RE | PORTING96 |
| APPENDE | | |
| | AND METHODS OF CONTRACEPTION | N100 |
| APPENDE | IX 5 STATIC PHYSICIAN'S GLOBAL ASSE | ESSMENT OF |
| | PSORIASIS (sPGA) | 104 |
| APPENDE | IX 6 PSORIASIS AREA AND SEVERITY IN | DEX (PASI)105 |
| APPENDI | | |
| | (CASPAR) | 113 |
| APPENDI | IX 17 JDA CRITERIA FOR SEVERITY ASSE | SSMENT OF |
| | PUSTULAR PSORIASIS (GENERALIZ) | ED PSORIASIS)118 |
| APPENDE | | |
| | (PASE) QUESTIONNAIRE | |
| APPENDE | | STIONNAIRE (PHQ-8)131 |
| APPENDE | IX 25 SUICIDAL IDEATION AND BEHAVIO DEFINITIONS | OR CATEGORIES AND132 |

## **LIST OF TABLES**

| Table 2: On Treatment Procedural Outline (IM011066): Week 0 through Week 20 | 16 | Table 1: Sc |
|---|---|---|
| Table 4: Study Treatments for Study Number | 0 | |
| · | | |
| Table 5: Selection and Timing of Dose | 49 | Table 4: St |
| | 49 | Table 5: Se |
| | 4 | Table 5: Se |

# **LIST OF FIGURES**

No table of figures entries found.

#### 1 PROTOCOL SUMMARY

## 1.1 Synopsis

**Protocol Title:** An Open-Label, Single-Arm, Multi-Center, Phase 3 Study to Evaluate the Efficacy and Safety of BMS-986165 in Japanese Subjects with Moderate-to-Severe Psoriasis

**Short Title:** Efficacy and Safety of BMS-986165 in Subjects with Moderate-to-Severe Psoriasis

**Study Phase: 3** 

### **Rationale:**

BMS-986165 is being evaluated as a therapeutic option for the treatment of subjects with moderate-to-severe plaque psoriasis based on results of a recently completed 12-week, randomized Phase 2, placebo-controlled, parallel-group study (Study IM011011). The Phase 2 study was conducted with the following 5 different BMS-986165 treatment arms: 3 mg every other day (QOD); 3 mg once daily (QD); 3 mg twice daily (BID); 6 mg BID; and 12 mg QD.

Overall, 267 subjects were randomized (44 to 45 subjects per treatment arm) in the Phase 2 study. All BMS-986165 treatment groups, except 3 mg QOD, achieved the primary endpoint of superiority compared with placebo in the proportion of subjects experiencing at least a 75% improvement in the Psoriasis Area and Severity Index (PASI 75) after 12 weeks of treatment. Compared with the placebo treatment group (6.7%), 38.6% (P = 0.0003), 68.9% (P < 0.0001), 66.7% (P < 0.0001) and 75% (P < 0.0001) of the subjects treated with BMS-986165 at 3 mg QD, 3 mg BID, 6 mg BID and 12 mg QD doses, respectively, achieved a PASI 75 response. The PASI 75 responses plateaued at a dose of 3 mg BID. The dose selected (6 mg QD) for the current global Phase 3 studies is expected to demonstrate equivalent efficacy to the 3 mg BID dose.

This open-label study (IM011066) being conducted in Japan is a supplement to the global Phase 3 study (IM011046) which is designed to confirm the efficacy and safety of BMS-986165 in a larger global population of subjects with moderate-to-severe plaque psoriasis. For approval in Japan, safety data collected from approximately 100 subjects dosed with BMS-986165 is needed. To achieve this: the IM011046 study is targeting to randomize approximately 52 Japanese subjects of which approximately 26 subjects will be dosed with BMS-986165; the IM011066 study is targeting to enroll and dose approximately 80 Japanese subjects.

In addition to subjects with plaque psoriasis, subjects with erythrodermic psoriasis and generalized pustular psoriasis will be allowed to enter the open-label study to explore the safety and efficacy in those rare variants of psoriasis for whom additional treatment options are limited. The open-label study design allows subjects with erythrodermic psoriasis and generalized pustular psoriasis to receive active treatment during the entire duration of the study as it would be unethical to have those subjects with these severe variants of psoriasis to receive placebo. To ensure the safety of these subjects, certain concomitant medications will be allowed at the time points defined per protocol.

### **Study Population:**

Japanese men and women  $\geq 20$  years of age:

- 1. Diagnosed with stable (defined as no morphology changes or significant flares of disease activity in the opinion of the investigator) plaque psoriasis for  $\geq 6$  months.
  - NOTE: Subjects with plaque psoriasis can also be classified to have psoriatic arthritis confirmed by Classification Criteria for Psoriatic Arthritis (CASPAR) (APPENDIX 13).
- 2. Having moderate-to-severe disease by involvement of ≥10% of body surface area (BSA) at both Screening Visit and Day 1, static Physician's Global Assessment (sPGA) ≥3 at both Screening Visit and Day 1, and PASI score ≥12 at both Screening Visit and Day 1.
- 3. Who are candidates for phototherapy or systemic therapy.
- 4. For generalized pustular psoriasis, those with prior history of or newly diagnosed generalized pustular psoriasis based on Japanese Dermatological Association (JDA)¹ criteria and have been on a stable treatment regimen for at least 2 weeks prior to Day 1; have erythematous lesions pustules involving ≥ 10% of body surface area (ie, score of at least 2 on the evaluation of skin symptoms [APPENDIX 17]) at both Screening Visit and Day 1; have a total JDA severity index score <14 (APPENDIX 17) at Screening Visit; and who are candidates for phototherapy or systemic therapy.
- 5. For erythrodermic psoriasis, involving ≥80% of BSA at screening and Day 1, who also have a history of plaque psoriasis, and who are candidates for phototherapy or systemic therapy.

### **Objectives and Endpoints:**

The objective of the study is to assess safety and efficacy of BMS-986165 6 mg QD in subjects with stable moderate-to-severe plaque psoriasis (with or without psoriatic arthritis), erythrodermic psoriasis, or generalized pustular psoriasis.

The primary endpoints are:

- sPGA 0/1 response assessed as a proportion of subjects with a sPGA score of 0 or 1 at Week 16
- PASI 75 response assessed as a proportion of subjects who achieve a 75% improvement from baseline in the PASI score at Week 16

The additional endpoints can be found in Section 3.

### **Overall Design:**

This will be a 52-week, multi-center, open-label, single-arm, Phase 3 study in approximately 80 Japanese subjects with moderate-to-severe stable, plaque psoriasis, generalized pustular psoriasis, or erythrodermic psoriasis. Subjects will undergo screening evaluations to determine eligibility within 28 days prior to administration of study medication. Following the screening process, approximately 80 qualified subjects will receive BMS-986165 6 mg QD for up to 52 weeks.

Enrollment should not occur until at least 8 days after the Screening Visit

A subject with at Week 24 may be treated with restricted topical medications, such as topical ultra-high to moderate potency corticosteroids (World Health Organization [WHO] Classes I-V), only at this time point at the discretion of the investigator.

Subjects who discontinue study treatment early are expected to remain in the study for continued follow-up until Week 52. Those completing 52 weeks of treatment may be eligible to roll over to a long-term extension study and be treated with BMS-986165 6 mg QD.

Note: Enrollment into the study will be divided into 2 enrollment periods: Parts A and B.

Part A will only enroll subjects diagnosed with generalized pustular psoriasis (~10 subjects) or erythrodermic psoriasis (~10 subjects). Part B will only enroll subjects diagnosed with plaque psoriasis (~60 subjects). Part A enrollment will begin at the initiation of IM011066. Part B enrollment will begin only after the targeted number of Japanese subjects (~52 subjects) have been randomized into the IM011046 study. Part A enrollment may continue once Part B enrollment has begun.

#### **Treatment Arms and Duration:**

Study treatment: Single-Arm BMS-986165 6 mg QD for 52 weeks

| | Study Drug for IM011066 | |
|-------------------|-------------------------|-----------|
| Medication | Potency | IP/Non-IP |
| BMS-986165 tablet | 6 mg | IP |

IP = investigational product

#### **Statistical Methods:**



### **General Methodology:**

As this is a single-arm study, no statistical tests for treatment comparisons will be conducted. All binary efficacy endpoints will be summarized using counts and percentages of subjects and all continuous efficacy endpoints will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, and maximum). Summaries will be provided for plaque psoriasis (including psoriatic arthritis), generalized pustular psoriasis, or erythrodermic psoriasis subjects separately.

#### **Safety Analysis:**

Treatment-emergent AEs and SAEs will be summarized using counts and percentages of subjects experiencing the event as well as the number of events by system organ class, preferred term, and treatment group. Vital signs, clinical laboratory test results, and ECG test results will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, and maximum) for continuous variables and frequency distributions (counts and percentages) for categorical variables.

## 1.2 Schedule of Activities (SOA)

The schedules of assessments and procedures are documented in Table 1 for screening, Table 2 for baseline through Week 20, and Table 3 for Week 24 through Week 52.

Table 1: Screening Procedural Outline (IM011066)

| Procedure | Screening<br>V1 | PsA Classification<br>Visit <sup>a</sup><br>V1A | Notes |
|---|---|---|---|
| <b>Eligibility Assessments</b> | | | |
| Informed Consent | X | | A subject is considered enrolled only when a protocol-specific informed consent is signed |
| Enroll Subject | X | | Obtain number from IRT |
| Inclusion/Exclusion Criteria | X | | Includes duration of plaque, erythrodermic, or generalized pustular psoriasis and documentation of presence of the type of psoriasis by the investigator |
| Medical History | X | | See Section 5.2 for complete eligibility criteria associated with medical history. Of note, subjects need to be screened for any current uncontrolled neuropsychiatric illness or history of suicidality; any history of TB; any congenital or acquired immunodeficiency; any significant drug allergy such as anaphylaxis; any cancer currently or in the previous 5 years. Investigators are encouraged to check whether subjects have had preventive health measures such as cancer screening (eg Pap smear, colonoscopy, mammograms) that is up-to-date according to local guidelines. |
| History of Tobacco Use | X | | Include description of current tobacco use |
| Psoriasis-related History | X | | Includes scalp symptoms, psoriatic arthritis/joint pain, nail involvement, palmoplantar involvement, genital involvement, history of other forms of psoriasis (eg, generalized pustular psoriasis, erythrodermic psoriasis) |
| Psoriasis-related Systemic Treatment | X | | History of: conventional systemic (eg, methotrexate), biologic, and/or phototherapy. For each therapy, include length of time on treatment and reason(s) for discontinuation (eg lack of efficacy, intolerance, side effects, loss of access to treatment) if applicable. |
| Psoriatic arthritis-related History | | $X^a$ | Includes history or presence of swollen joints/digits, joint pain, entheseal pain, and/or morning stiffness. |
| Psoriatic arthritis classification based on CASPAR criteria | | $X^a$ | Subjects with a medical history of psoriatic arthritis or who report symptoms of psoriatic arthritis with a PASE questionnaire score of ≥47, will undergo confirmation of their classification of psoriatic arthritis by the CASPAR criteria. For the CASPAR Criteria, historical rheumatoid factor results, and historical hand or foot radiograph results are acceptable. |

Table 1: Screening Procedural Outline (IM011066)

| Procedure | Screening<br>V1 | PsA Classification<br>Visit <sup>a</sup><br>V1A | Notes |
|---|---|---|---|
| Assessment of GPP severity using JDA criteria (ie, skin symptoms, systemic symptoms and laboratory findings) <sup>b</sup> | X | | See APPENDIX 17 |
| Other Prior and Concomitant Treatments | X | | Includes topical treatments and shampoos for psoriasis and all medications for other conditions such as cardiovascular and mood disorders. |
| Safety Assessments | | | |
| Physical Examination (PE) | X | | Complete PE |
| Physical Measurements | X | | Includes height and weight |
| Vital Signs | X | | Includes (ear or oral) body temperature, respiratory rate, seated blood pressure and heart rate. Blood pressure and heart rate should be measured after the subject has been resting quietly for at least 5 minutes. |
| Electrocardiogram (ECG) | X | | ECGs should be recorded after the subject has been supine for at least 5 minutes. |
| Chest Imaging (eg, Chest x-ray) | X | | Chest imaging is required if not performed within 6 months of Screening Visit, copy of radiology report must be on file and reviewed by PI. Section 8.4.4 |
| Neuropsychiatric Illness Assessment | X | | Based on subject/family response, medical history/medical records, investigator judgment |
| PHQ-8 | X | | For establishing baseline depression severity |
| Suicidal Ideation and Behavior<br>Assessment | X | | Based on subject/family response, medical history/medical records, investigator judgment |
| eC-SSRS | X | | eC-SSRS Assessment: Response of "Actual Suicide Attempt-Lifetime" or suicidal ideation (Severity of 4 or 5) or suicidal behavior will be exclusionary. Rescreening will not be allowed. Section 8.4.7 |
| Monitor for Serious Adverse Events | X | | All SAEs must be collected from the date of subject's written consent until 30 days post discontinuation of dosing or subject's participation in the study. |
| <b>Laboratory Tests</b> | | | |
| Hematology | X | | Complete Blood Count (CBC) with differential |
| Chemistry Panel | X | | |

Table 1: Screening Procedural Outline (IM011066)

| Procedure | Screening<br>V1 | PsA Classification<br>Visit <sup>a</sup><br>V1A | Notes |
|---|---|---|---|
| Lipid Panel | X | | |
| Urinalysis | X | | |
| Hemoglobin A1C | X | | |
| TSH | X | | If TSH above normal reference range, test free T4; if TSH below normal range, test free T4 & T3 |
| Serology | X | | Includes HCV antibody, HBsAg, HBsAb, HBcAb, HBV DNA, and HIV antibodies |
| Tuberculosis Test | X | | In accordance with QuantiFERON®-TB Gold. (details are described in Section 8.4.4). |
| Pregnancy Test (serum) | X | | For WOCBP only |
| Follicle Stimulating Hormone (FSH) | X | | To confirm menopausal status (see APPENDIX 4) |
| (1→3)-beta-D glucan | X | | |
| Clinical Efficacy/Health Outcomes | | | |
| sPGA | X | | |
| PASI | X | | |
| BSA | X | | |
| PASE Questionnaire | X | | For subjects with psoriatic arthritis type complaints to screen for presence of psoriatic arthritis |

BSA = body surface area; CASPAR = Classification Criteria for Psoriatic Arthritis; CBC = complete blood count; DNA = deoxyribonucleic acid; ECG = electrocardiogram; eC-SSRS = electronic Columbia-Suicide Severity Rating Scale; FSH = follicle-stimulating hormone; GPP = generalized pustular psoriasis; HBV = hepatitis B virus; HBcAb = hepatitis B surface antibody; HBsAb = hep

IRT = interactive response technology; PASE = psoriatic arthritis screening and evaluation; PASI = Psoriasis Area and Severity Index; PE = physical examination;

PHQ-8 = eight-item Patient Health Questionnaire; PI = principal investigator; PsA = psoriatic arthritis; SAE = serious adverse events; sPGA = static Physician Global Assessment; T3 = triiodothyronine; T4 = thyroxine; TB = tuberculosis; TSH = thyroid-stimulating hormone; V = visit; WOCBP = women of childbearing potential

<sup>a</sup>Visit 1A applies to subjects only with a medical history of psoriatic arthritis (PsA) or suspected to have symptoms of PsA. This visit is needed only if PsA assessments can't be completed at Visit 1. If the visit is needed, it must occur prior to the baseline visit (Visit 2). See Section 4.1.1 for more details.

<sup>b</sup>Only in subjects with generalized pustular psoriasis

Table 2: On Treatment Procedural Outline (IM011066): Week 0 through Week 20

| Clinical Efficacy/Health Outcomes SPGA X X X X X X X X X X X X X X X X X X X | Procedure | Week 0<br>Baseline/<br>D1<br>V2 | Week 1<br>D8<br>(±3 d)<br>V3 | Week 2<br>D15<br>(±3 d)<br>V4 | Week 4<br>D29<br>(±3 d)<br>V5 | Week 8<br>D57<br>(±3 d)<br>V6 | Week 12<br>D85<br>(±3 d)<br>V7 | Week 16<br>D113<br>(±3 d)<br>V8 | Week 20<br>D141<br>(±3 d)<br>V9 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| | Clinical Efficacy/Health Outcomes | | | | | | | | | |
| | | 71 | 71 | 71 | 71 | 71 | 71 | 71 | | |

Table 2: On Treatment Procedural Outline (IM011066): Week 0 through Week 20

| Procedure | Week 0<br>Baseline/<br>D1<br>V2 | Week 1<br>D8<br>(±3 d)<br>V3 | Week 2<br>D15<br>(±3 d)<br>V4 | Week 4<br>D29<br>(±3 d)<br>V5 | Week 8<br>D57<br>(±3 d)<br>V6 | Week 12<br>D85<br>(±3 d)<br>V7 | Week 16<br>D113<br>(±3 d)<br>V8 | Week 20<br>D141<br>(±3 d)<br>V9 | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Sector Assessment | | | | | | | | | |
| Safety Assessments Complete PE | X | | | | | | X | | |
| Targeted PE | | X | X | X | X | X | | X | See Section<br>8.4.1 |
| Body Weight | X | | | | X | | X | | |
| Vital Signs | X | X | X | X | X | X | X | X | |
| Electrocardiogram (ECG) | X | | | | | | X | | |
| PHQ-8 | X | | | | X | | X | | See Section<br>8.4.6.1 |
| eC-SSRS Assessment | X | | | | X | | X | | Suicidal<br>Ideation and |

Table 2: On Treatment Procedural Outline (IM011066): Week 0 through Week 20

| Procedure | Week 0<br>Baseline/<br>D1<br>V2 | Week 1<br>D8<br>(±3 d)<br>V3 | Week 2<br>D15<br>(±3 d)<br>V4 | Week 4<br>D29<br>(±3 d)<br>V5 | Week 8<br>D57<br>(±3 d)<br>V6 | Week 12<br>D85<br>(±3 d)<br>V7 | Week 16<br>D113<br>(±3 d)<br>V8 | Week 20<br>D141<br>(±3 d)<br>V9 | Notes |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Behavior since last visit |
| Adverse Event Assessment | X | X | X | X | X | X | X | X | |
| Concomitant Medication Use | X | X | X | X | X | X | X | X | |
| <b>Laboratory Tests</b> | | | | | | | | | |
| Hematology | X | X | X | X | X | X | X | X | |
| Lymphocyte Subsets (TBNK) | X | | | | X | | X | | |
| Chemistry Panel | X | X | X | X | X | X | X | X | If CK >2.5 x<br>ULN, reflex<br>testing is<br>required (See<br>Section 8.4.5) |
| Hemoglobin A1C | X | | | | | | X | | |
| Fasting Lipid Panel | X | | | | X | | X | | |
| Fasting Plasma Glucose | X | | | | X | | X | | |
| Urinalysis | X | | | | | | X | | |
| Serum Immunoglobulin Levels<br>(IgM, IgG, IgA, IgE) | X | | | | X | | X | | |
| Pregnancy Test (Urine) | X | | | X | X | X | X | X | WOCBP only |
| HBV DNA Test <sup>h</sup> | X | | | X | X | X | X | X | |

Table 2: On Treatment Procedural Outline (IM011066): Week 0 through Week 20

| Procedure | Week 0<br>Baseline/<br>D1<br>V2 | Week 1<br>D8<br>(±3 d)<br>V3 | Week 2<br>D15<br>(±3 d)<br>V4 | Week 4<br>D29<br>(±3 d)<br>V5 | Week 8<br>D57<br>(±3 d)<br>V6 | Week 12<br>D85<br>(±3 d)<br>V7 | Week 16<br>D113<br>(±3 d)<br>V8 | Week 20<br>D141<br>(±3 d)<br>V9 | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Study Treatment | | | | | | | | | |
| Enrollment | X | | | | | | | | |
| Dispense Study Treatment | X | | X | X | X | X | X | X | |
| Study Treatment Compliance | | X | X | X | X | X | X | X | See Section 6.6 |

Table 2: On Treatment Procedural Outline (IM011066): Week 0 through Week 20

| Procedure | Week 0<br>Baseline/<br>D1<br>V2 | Week 1<br>D8<br>(±3 d)<br>V3 | Week 2<br>D15<br>(±3 d)<br>V4 | Week 4<br>D29<br>(±3 d)<br>V5 | Week 8<br>D57<br>(±3 d)<br>V6 | Week 12<br>D85<br>(±3 d)<br>V7 | Week 16<br>D113<br>(±3 d)<br>V8 | Week 20<br>D141<br>(±3 d)<br>V9 | Notes |
|---|---|---|---|---|---|---|---|---|---|
| ACR = American College of Rheuma | ntology: | | CA | SPAR = Cla | ssification Cri | teria for Psor | iatic Arthritis: | CK = creatir | ne kinase: |
| D = Day; d = days; | ,,,,, | | | | | | | | RS = electronic |
| Columbia-Suicide Severity Rating Sca | le; | | | | | | | | |
| | | | | | | | | HBV = hepa | titis B virus; |
| DACI — D | _ | nunoglobulir | - | | | | | | |
| PASI = Psoriasis Area and Severity In<br>PHQ-8 = eight-item Patient Health Que | | ysicai exami | nation; | | | | | | |
| 1110 0 eight teim rutent freath Que | stronnane, | S | PGA = static 1 | Physician Glo | bal Assessmen | ıt; | | | |
| TBNK = T cells, B cells, and natural ki | ller cells; UL | | | | | | = Week; WO | CBP = women | of childbearing |
| potential | | | | | | | | | |

gIf sample is missed, it may be taken at any visit once informed consent is obtained

<sup>h</sup>Testing for HBV DNA will occur every 4 weeks for subjects who are negative HBsAg, but positive HBsAb and/or positive HBcAb with Hepatitis B virus DNA <2.1 log copies/mL [20IU/mL] at screening.

When multiple assessments are conducted at a single visit, the following is the order in which they should be done:

- 1) Health outcomes assessments
- 2)Safety assessments (eg, vitals, AEs)
- 3)Clinical efficacy assessments
- 4)Laboratory tests (eg, safety laboratory tests,

On fasting days, safety assessments can be done first followed by blood draws, and then health outcomes and finally efficacy assessments. The dose of the drug on a visit day is to be taken after blood draws.

Table 3: On Treatment Procedural Outline (IM011066): Week 24 Through Week 52

| Procedure | Week 24<br>D169<br>(±3 d)<br>V10 | Week 28<br>D197<br>(±3 d)<br>V11 | Week 32<br>D225<br>(±3 d)<br>V12 | Week 36<br>D253<br>(±3 d)<br>V13 | Week 40<br>D281<br>(±3 d)<br>V14 | Week 44<br>D309<br>(±3 d)<br>V15 | Week 48<br>D337<br>(±3 d)<br>V16 | Week 52 <sup>a</sup><br>(or early<br>DC)<br>D365<br>(±3 d)<br>V17 | Safety<br>Follow-Up <sup>b</sup><br>(Week 56)<br>D393<br>(±3 d)<br>V18 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|

Table 3: On Treatment Procedural Outline (IM011066): Week 24 Through Week 52

| Procedure | Week 24<br>D169<br>(±3 d)<br>V10 | Week 28<br>D197<br>(±3 d)<br>V11 | Week 32<br>D225<br>(±3 d)<br>V12 | Week 36<br>D253<br>(±3 d)<br>V13 | Week 40<br>D281<br>(±3 d)<br>V14 | Week 44<br>D309<br>(±3 d)<br>V15 | Week 48<br>D337<br>(±3 d)<br>V16 | Week 52 <sup>a</sup><br>(or early<br>DC)<br>D365<br>(±3 d)<br>V17 | Safety<br>Follow-Up <sup>b</sup><br>(Week 56)<br>D393<br>(±3 d)<br>V18 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Safety Assessments | | | | | | | | | | |
| Full Physical Examination | X | | | | | | | X | X | |
| Targeted Physical<br>Examination | | X | X | X | X | X | X | | | |
| Body Weight | X | | | X | | | | X | X | |
| Vital Signs | X | X | X | X | X | X | X | X | X | |
| Electrocardiogram | X | | | | | | | X | | |
| PHQ-8 | | X | | | X | | | X | | See Section 8.4.6.1 |
| eC-SSRS | | X | | | X | | | X | | Suicidal Ideation and<br>Behavior since last visit |
| Adverse Event Assessment | X | X | X | X | X | X | X | X | X | |
| Concomitant Medication<br>Use | X | X | X | X | X | X | X | X | X | |

Table 3: On Treatment Procedural Outline (IM011066): Week 24 Through Week 52

| Procedure | Week 24<br>D169<br>(±3 d)<br>V10 | Week 28<br>D197<br>(±3 d)<br>V11 | Week 32<br>D225<br>(±3 d)<br>V12 | Week 36<br>D253<br>(±3 d)<br>V13 | Week 40<br>D281<br>(±3 d)<br>V14 | Week 44<br>D309<br>(±3 d)<br>V15 | Week 48<br>D337<br>(±3 d)<br>V16 | Week 52 <sup>a</sup><br>(or early<br>DC)<br>D365<br>(±3 d)<br>V17 | Safety<br>Follow-Up <sup>b</sup><br>(Week 56)<br>D393<br>(±3 d)<br>V18 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| <b>Laboratory Tests</b> | | | | | | | | | | |
| Hematology | X | X | X | X | X | X | X | X | X | |
| Lymphocyte Subsets (TBNK) | | | | X | | | | X | | |
| Chemistry Panel | X | X | X | X | X | X | X | X | X | If CK > 2.5 x ULN,<br>reflex testing is required<br>(see Section 8.4.5) |
| Fasting Lipid Panel | X | | | | | | | X | | |
| Fasting Plasma Glucose | X | | | | | | | X | | |
| Hemoglobin A1C | | | | X | | | | X | | |
| Urinalysis | | | | X | | | | X | X | |
| Serum Immunoglobulin<br>Levels (IgM, IgG, IgA, IgE) | | | | X | | | | X | | |
| Pregnancy Test (Urine) | X | X | X | X | X | X | X | X | X | WOCBP only |
| HBV DNA Test <sup>i</sup> | X | X | X | X | X | X | X | X | X | |

| Table 3: O | n Treatme | nt Procedu | ral Outline | (IM011066) | : Week 24 | Through W | eek 52 | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Week 24<br>D169<br>(±3 d)<br>V10 | Week 28<br>D197<br>(±3 d)<br>V11 | Week 32<br>D225<br>(±3 d)<br>V12 | Week 36<br>D253<br>(±3 d)<br>V13 | Week 40<br>D281<br>(±3 d)<br>V14 | Week 44<br>D309<br>(±3 d)<br>V15 | Week 48<br>D337<br>(±3 d)<br>V16 | Week 52 <sup>a</sup><br>(or early<br>DC)<br>D365<br>(±3 d)<br>V17 | Safety<br>Follow-Up <sup>b</sup><br>(Week 56)<br>D393<br>(±3 d)<br>V18 | Notes |
| <b>Study Treatment</b> | | | | | | | | | | |
| Dispense Study Treatment | X | X | X | X | X | X | X | | | |
| Study Treatment<br>Compliance | X | X | X | X | X | X | X | X | | |
| ACR = American College of 1<br>= Day; d = days; | Rheumatology | | | CASPAR = Cla<br>yribonucleic ac | | | | | | D<br>Severity Rating |
| Scale; immunoglobulin; | | | | | HBV = | hepatitis B v | irus; | | | Ig = PE = physical |
| examination; | | | | | | PH | IQ-8 = eight | item Patient | Health Questic | onnaire; |

TBNK = T cells, B cells, and natural killer cells; ULN = upper limit of normal; V = visit; ; Wk = Week; WOCBP = women of childbearing potential

<sup>a</sup>For subjects who discontinue treatment prior to Week 52, please refer to Section 7.1 for more details.

<sup>b</sup>For subjects who do not continue in a long-term extension study

<sup>i</sup>Testing for HBV DNA will occur every 4 weeks for subjects who are negative HBsAg, but positive HBsAb and/or positive HBcAb with Hepatitis B virus DNA <2.1 log copies/mL [20IU/mL] at screening.

When multiple assessments are conducted at a single visit, the following is the recommended order in which they should be done:

- 1) Health outcomes assessments
- 2) Safety assessments (eg, vitals, AEs)
- 3) Clinical efficacy assessments
- 4) Laboratory tests (eg, safety laboratory tests,

On fasting days, safety assessments can be done first followed by blood draws, and then health outcomes and finally efficacy assessments.

The dose of the drug on a visit day is to be taken after blood draws.

#### STUDY ACKNOWLEDGMENT/DISCLOSURE

I understand that this protocol contains information that is confidential and proprietary to Bristol-Myers Squibb Company (BMS). Any supplemental information that may be added to this document is also confidential and proprietary to BMS and must be kept in confidence in the same manner as the contents of this protocol.

I have read the original protocol/revised protocol and agree that it contains all necessary details for carrying out the study as described. I will conduct this protocol as outlined therein and will make a reasonable effort to complete the study within the time designated.

I will provide copies of the protocol and access to all information furnished by BMS to study personnel under my supervision. I will discuss this material with them to ensure that they are fully informed about the investigational product and the study.

I will provide protocol information to my Institutional Review Board(s) [IRB(s)] or Independent Ethics Committee(s) [IEC(s]. I understand that original protocol/revised protocols must be reviewed by the Institutional Review Board or Independent Ethics Committee overseeing the conduct of the study and approved or given favorable opinion by all necessary health authorities before implementation unless to eliminate an immediate hazard to subjects.

I agree that the contents of the protocol may not be disclosed to any other person or entity or used for any other purpose without the prior written consent of BMS. The foregoing shall not apply to disclosure required by governmental regulations or laws; however, I will give prompt notice to BMS of any such disclosure.

I agree that the study data derived from this protocol may only be used and disclosed in furtherance of the protocol, for the medical treatment of a study subject or for publication of study results in accordance with the terms of the clinical trial agreement or as otherwise permitted by the terms of the clinical trial agreement.

I agree not to collect or use samples (eg, tissue, blood, serum, urine) or collect data (other than for diagnostic or treatment purposes) from the study subjects while enrolled in the study, except as expressly permitted by the protocol or the terms of the clinical trial agreement.

I understand that I may terminate or suspend enrollment of the study at any time if it becomes necessary to protect the best interests of the study subjects. Unless otherwise provided in the clinical trial agreement, the study may be terminated at any time by BMS, with or without cause.

| Original Protocol: | Revised Protocol: |
|---------------------------------------------------|---------------------|
| Protocol Number: IM011066 Revised Protocol 04 | Site Number: |
| Date of Protocol or Revised Protocol: 07-May-2020 | |
| IND Number: 131,993 | EUDRACT Number: N/A |
| Investigator: | Date: |
| (signature) | |
| (printed name) | |

### 2 INTRODUCTION

Psoriasis is a chronic inflammatory skin disorder, characterized primarily by erythematous scaly plaques, that affects up to 3% of the general population. Men and women are equally affected and it can present at any age.<sup>2,3</sup> Several studies have observed a bimodal distribution of psoriasis onset with the first peak ranging from 15 to 22 years of age, and the second peak ranging from 55 to 60 years of age. 4-6 The most common form of psoriasis (58% to 97% of cases) is plaque psoriasis (psoriasis vulgaris), with less common forms being guttate, pustular, inverse (flexural), and erythrodermic psoriasis. The disease can have a fluctuating relapsing course, with flares that may be induced by factors such as infections, trauma, smoking, and stress<sup>4</sup> Psoriasis can involve skin in any part of the body; particularly disabling is the involvement of specific anatomic regions, such as hands and feet (palmoplantar), face, scalp, and nails. Disease severity can be classified by body surface area (BSA) involvement with mild defined as ≤ 10% BSA, and moderate-to-severe as > 10% BSA. Psoriasis has a profound impact on quality of life and can lead to psychological, social and economic consequences, especially in moderate-to-severe disease. This condition is also associated with an increased risk of depression, occurrence of sleep disturbances, social stigma and decreased work productivity. 8 Commonly associated comorbidities found in psoriasis patients include diabetes mellitus and metabolic syndrome. In patients with more severe forms of the disease, life expectancy is decreased due to an increase of cardiovascular risk.9

Treatments include topical preparations, eg, corticosteroids, vitamin D analogs, calcineurin inhibitors, and salicylic acid; phototherapy modalities, including PUVA (psoralens with ultraviolet A) and narrow band ultraviolet B (UVB); and systemic therapies. In moderate-to-severe disease, systemic treatments are usually needed and may include oral agents (retinoids, methotrexate, cyclosporine, and apremilast) or injectables (eg, biologics such as tumor necrosis factor (TNF) inhibitors etanercept, infliximab, and adalimumab) anti- interleukin (IL)-12/23p40 antibody (ustekinumab), IL-17 antagonists (secukinumab, ixekizumab, brodalumab), and anti-IL-23p19 antibody (guselkumab). Many of these treatments are associated with increased risk of AEs such as hepatotoxicity and neutropenia (methotrexate); nephrotoxicity (cyclosporine); depression and weight loss (apremilast); serious infections (cytokine inhibitors); and candidiasis and Crohn's disease (IL-17 antagonists).

Although effective therapeutic options are available, under-treatment or nontreatment of psoriasis has been reported in up to half of surveyed patients (based on absence of treatment and/or dissatisfaction with treatment). Many patients with severe disease are still being managed with only topicals therapies, and patients consider many of the treatments to be inadequate. Accordingly, there remains a need for more effective oral options, when compared with currently available agents, that would improve efficacy responses and increase adherence to treatment.

## 2.1 Study Rationale

BMS-986165 is being evaluated as a therapeutic option for the treatment of subjects with moderate-to-severe plaque psoriasis based on results of a recently completed 12-week randomized Phase 2, placebo-controlled, parallel-group study with 5 different BMS-986165 treatment arms: 3 mg QOD; 3 mg QD; 3 mg BID; 6 mg BID; and 12 mg QD (Study IM011011). Overall,

267 subjects were randomized (44 to 45 subjects per treatment arm) in the Phase 2 study. All BMS-986165 treatment groups, except 3 mg QOD, achieved the primary endpoint of superiority compared with placebo in the proportion of subjects achieving at least a 75% improvement in the Psoriasis Area and Severity Index (PASI 75) after 12 weeks of treatment. Compared with placebo treatment group, in which 6.7% of the subjects achieved PASI 75 response, 38.6% (P = 0.0003), 68.9% (P < 0.0001), 66.7% (P < 0.0001) and 75% (P < 0.0001) of subjects treated with 3 mg QD, 3 mg BID, 6 mg BID and 12 mg QD achieved PASI 75, respectively. The PASI 75 responses plateaued at a dose of 3 mg BID, and the Phase 3 dose selected (6 mg QD) is expected to demonstrate equivalent efficacy to the 3 mg BID dose.

Also, there was a clinically significant proportion of subjects treated with BMS-986165 achieving an sPGA score of 0 or 1 compared with placebo at Week 12. Compared with the placebo treatment group in which 6.7% of the subjects achieved an sPGA score of 0 or 1, 41.5%, 75.6%, 65.9%, and 75% of the subjects treated with 3 mg QD, 3 mg BID, 6 mg BID and 12 mg QD achieved an sPGA score of 0 or 1, respectively.<sup>20</sup>

This open-label study (IM011066) being conducted in Japan is a supplement to the global Phase 3 study (IM011046) which is designed to confirm the efficacy and safety of BMS-986165 in a larger global population of subjects with moderate-to-severe plaque psoriasis. For approval, Japan requires safety data collected on approximately 100 subjects who receive BMS-986165. To achieve this number, this open-label study is expected to enroll approximately 80 Japanese subjects and the global study is expected to enroll approximately 52 Japanese subjects of which approximately 26 subjects will be dosed with BMS-986165 from Day 1.

In addition to subjects with plaque psoriasis, subjects with erythrodermic psoriasis and generalized pustular psoriasis will be allowed to enter the open-label study to explore the safety and efficacy in those rare variants of psoriasis, for whom additional treatment options are limited. The open-label study design allows subjects with erythrodermic psoriasis and generalized pustular psoriasis to receive active treatment during the entire duration of the study as it would be unethical to have those subjects with severe variants of psoriasis receive placebo. To ensure the safety of these subjects, certain concomitant medications will be allowed at the time points defined per protocol.

## 2.2 Background

Tyrosine kinase 2 (TYK2) is a nonreceptor tyrosine kinase associated with receptors for the p40-containing cytokines IL-12 and IL-23, as well as the Type I interferon (IFN) receptor, and is required for the activation of downstream signaling pathways. TYK2 catalyzes the phosphorylation of the intracellular receptor domains and signal transducer and activator of transcription (STAT) proteins resulting in the activation of STAT-dependent transcription and functional responses specific for these cytokines. Peculose TYK2-dependent cytokines (eg, Type I IFNs, IL-12, IL-23) are distinct from those dependent on closely related Janus kinase (JAK) family members JAK1/JAK3 (eg, IL-2, IL-15, IL-7) or JAK2 (eg, erythropoietin, thrombopoietin, GM-CSF), a TYK2 Inhibitor would be expected to have a highly differentiated profile from inhibitors of other JAK family kinases. TYK2-dependent pathways and the cytokine networks they modulate (eg IL-23/IL-17, IFNα) have been implicated in the pathophysiology of multiple immune-mediated diseases, including psoriasis, lupus, spondyloarthritides, and Crohn's disease.

BMS-986165 is a potent, highly selective, oral, small molecule-inhibitor of TYK2. A comprehensive in vitro and in vivo characterization of BMS-986165 has been established and supports the development of this compound in humans. Inhibition of TYK2 is expected to provide therapeutic benefit for subjects with psoriasis for multiple reasons: 1) Many of the pathways in the TYK2 signaling cascade (IFNα, IL-12/IL-23 and the downstream mediators IL-17 and IL-22) have been implicated in pathogenesis of psoriasis<sup>5</sup> 2) Biologic agents targeting the IL-17, IL-23p19, and IL-12/23 p40 pathways have been approved and are highly efficacious in the treatment of psoriasis.

## 2.2.1 Early Clinical Development

The clinical data available to date supporting the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of BMS-986165 are from 5 completed Phase 1 studies in healthy subjects (IM011002, IM011015, IM011016, IM011031, and IM011039) and 1 completed Phase 2 study in adult subjects with moderate-to-severe plaque psoriasis (IM011011).

Overall, BMS-986165 has been generally well-tolerated across all studies, and no safety issues have been identified to limit the investigation of the dose of BMS-986165 up to 12 mg QD in further clinical studies. A detailed description of the chemistry, pharmacology, efficacy, and safety of BMS-986165 is provided in the Investigator Brochure (IB).





### 3 OBJECTIVES AND ENDPOINTS

The objective of the study is to assess safety and efficacy of BMS-986165 6 mg QD in subjects with stable moderate-to-severe plaque psoriasis (with or without psoriatic arthritis [PsA]), erythrodermic psoriasis, or generalized pustular psoriasis.

The primary endpoints are:

- sPGA 0/1 response assessed as a proportion of subjects with a sPGA score of 0 or 1 at Week 16
- PASI 75 response assessed as a proportion of subjects who achieve a 75% improvement from baseline in the PASI score at Week 16






#### 4 STUDY DESIGN

## 4.1 Overall Design

This will be a 52-week, multi-center, open-label, single-arm, Phase 3 study in approximately 80 Japanese subjects with moderate-to-severe stable, plaque psoriasis, generalized pustular psoriasis, or erythrodermic psoriasis.

The duration of study participation is approximately 60 weeks and will be divided into the following periods: screening (up to 4 weeks), treatment (52 weeks), and follow-up (4 weeks).

Physical examinations, 12-lead ECGs, clinical laboratory evaluations, and other assessments will be done at select visits during the study. Subjects in this study will be monitored for AEs.

Note: Enrollment into the study will be divided into 2 enrollment periods: Parts A and B.

Part A will only enroll subjects diagnosed with generalized pustular psoriasis (~10 subjects) or erythrodermic psoriasis (~10 subjects). Part B will only enroll subjects diagnosed with plaque psoriasis (~60 subjects). Part A enrollment will begin at the initiation of IM011066. Part B enrollment will begin only after the targeted number of Japanese subjects (~52 subjects) have been randomized into the IM011046 study. Part A enrollment may continue once Part B enrollment has begun.

# 4.1.1 Screening Period

Subjects will be evaluated during the screening period to ensure they meet eligibility criteria. A detailed medical history will be done at this time, as well as a complete physical examination. Psoriasis-related history, which will include length of diagnosis, body involvement, and history of systemic treatment, will be assessed here. Depression and suicidality assessments will also be performed. An evaluation for tuberculosis (TB) will be done based on medical history, recent chest imaging, and a QuantiFERON®-TB Gold test.

Subjects with a medical history of psoriatic arthritis or who report symptoms of psoriatic arthritis with a PASE questionnaire score of ≥47, will undergo confirmation of their classification of psoriatic arthritis by the Classification criteria for Psoriatic ARthritis (CASPAR) criteria (APPENDIX 13)

It is preferable that a rheumatologist classify PsA by CASPAR criteria and perform joint assessments in a subject who has a history of psoriatic arthritis or who is presenting with symptoms suggestive of PsA. If assistance from a rheumatologist is not possible at the site, then a

dermatologist who is trained by a rheumatologist can classify a subject by CASPAR criteria as having PsA and perform the joint assessments for the subject in the study.

If these assessments can't be completed at Visit 1, subjects may return to complete these assessments at Visit 1A which must occur prior to the baseline visit (Visit 2).

#### 4.1.2 Treatment Period

Qualified subjects who have completed the screening procedures and have met the inclusion/exclusion criteria will be enrolled on Day 1 to receive BMS-985165 6 mg QD. Additional details are provided in Section 6.1.

Enrollment should not occur until at least 8 days after the Screening Visit

#### 4.1.3 Week 16

The primary endpoints (sPGA 0/1 and PASI 75) will be assessed at Week 16.

#### 4.1.4 Week 24

During the Week 24 assessment, a subject who has an may be treated with restricted topicals/shampoos as described in Section 6.7.1 at the investigator's discretion. These treatments may be only initiated at Week 24, and not at subsequent time points. A subject who is initiated on these treatments at Week 24 may use them as needed per the investigator's judgment through Week 52.

## 4.1.5 Week 52 and Follow-up Period

The follow-up period is a 4-week window after the Week 52 visit, unless the subject rolls over into the long-term extension study. The subject will be encouraged to report any SAEs or AEs experienced during this time.

Subjects who discontinue study treatment early should remain in the study for protocol-specified procedures (please refer to Section 7.1 for more details).

Subjects completing 52 weeks of treatment may be eligible to roll over to a long-term extension study and be treated with BMS-986165 6 mg QD.

# 4.1.6 Data Monitoring Committee and Other External Committees

# 4.1.6.1 Infection Adjudication Committee

An independent Infection Adjudication Committee, composed of individuals with relevant expertise, will blindly review and adjudicate infection AEs, such as opportunistic infections, influenza, herpes zoster, and TB, reported in the study per criteria specified in a separate charter. Additional information about these infections may be collected on the case report form (CRF) in order to characterize and understand them. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee members will not be investigators on the study.

## 4.1.6.2 CV Adjudication Committee

An independent cardiovascular (CV) Adjudication Committee, composed of individuals with relevant expertise, will blindly review and adjudicate cardiovascular and cerebrovascular AEs such as, but not limited to, Major Adverse Cardiovascular Events (MACE) that include death, non-fatal myocardial infarction, non-fatal stroke; revascularization procedures; heart failure; dysrhythmias; heart blocks; and thrombotic events reported in the study per criteria specified in a separate charter. Additional information about cardiovascular and cerebrovascular AEs may be collected on the CRF in order to characterize and understand them. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee members will not be investigators on the study.

## 4.1.6.3 Suicidal Ideation and Behavior (SIB) Adjudication Committee

An independent Suicidal Ideation and Behavior Adjudication Committee, composed of individuals with relevant expertise, will blindly review and adjudicate suicidal ideation/behavior reported in the study per criteria specified in a separate charter. Additional information about suicidal ideation/behavior may be collected on the CRF. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee members will not be investigators on the study.

## 4.2 Number of Subjects

Approximately 80 qualified subjects will receive BMS-986165 6 mg QD. It is anticipated that, among these 80 subjects, there will be approximately 60 subjects with plaque psoriasis, approximately 10 subjects with generalized pustular psoriasis, and approximately 10 subjects with erythrodermic psoriasis.

# 4.3 End of Study Definition

The duration of study participation for individual subjects is expected to be up to 60 weeks (420 days), which includes screening (up to 4 weeks), treatment (52 weeks) and follow-up (up to 4 weeks) periods.

The start of the study is defined as the first visit for the first subject screened. The end of the study is defined as the last visit or scheduled procedure shown in the Schedule of Activities (Section 1.2) for the last subject. Study completion is defined as the final date on which data were or are expected to be collected (Week 56 for collection of potential SAEs).

# 4.4 Scientific Rationale for Study Design

This open-label, Phase 3 study will be conducted in Japanese subjects with moderate-to-severe psoriasis who are candidates for systemic psoriasis therapy This study is a supplement to the Phase 3 study (IM011046) designed to confirm the efficacy and safety of BMS-986165 compared with placebo and apremilast in a larger global population of subjects with moderate-to-severe plaque psoriasis that will include around 52 Japanese subjects with 26 dosed from Day 1 with BMS-986165 in a blinded manner. This study will closely mimic the global study and will evaluate

the subjects achieving sPGA of 0/1 and PASI 75 at Week 16, which are standard measures of efficacy in clinical trials of psoriasis treatments.

For approval in Japan, safety data collected from approximately 100 subjects dosed with BMS-986165 is needed. To achieve this: the IM011046 study is targeting to randomize approximately 52 Japanese subjects of which approximately 26 subjects will be dosed with BMS-986165; the IM011066 study is targeting to enroll and dose approximately 80 Japanese subjects. In addition to subjects with plaque psoriasis, subjects with erythrodermic psoriasis and generalized pustular psoriasis will also be allowed to enter the open-label study to explore the safety and efficacy in those rare variants of psoriasis, for whom additional treatment options are limited. The open-label study design allows subjects with erythrodermic psoriasis and generalized pustular psoriasis to receive active treatment during the entire duration of the study as it would be unethical to have those subjects with severe variants of psoriasis receive placebo. To ensure the safety of these subjects, certain concomitant medications will be allowed at the time points defined per protocol.



#### 5 STUDY POPULATION

Eligibility criteria for this study have been carefully considered to ensure 1) selection of appropriate subjects with psoriasis, 2) safety of the study subjects and 3) the results of the study can be used for regulatory filing and other purposes. It is imperative that subjects fully meet all eligibility criteria.

All screening and enrollment evaluations must be completed and reviewed to confirm that potential subjects meet all eligibility criteria. The investigator will maintain a screening log to record details of all subjects screened and to confirm eligibility or record reasons for screening failure, as applicable.

#### 5.1 Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

## 1) Signed Written Informed Consent

a) Subjects must be willing to participate in the study and sign the informed consent form (ICF)

## 2) Type of Subject and Target Disease Characteristics

- a) For subjects with plaque psoriasis:
  - i) Men and women diagnosed with stable plaque psoriasis for 6 months or more. Stable plaque psoriasis is defined as no morphology changes or significant flares of disease activity in the opinion of the investigator
  - ii) Deemed by the investigator to be a candidate for phototherapy or systemic therapy
  - iii) ≥10% of BSA involvement at both Screening Visit and Day 1
  - iv) PASI score ≥12, sPGA ≥3 at both Screening Visit and Day 1 NOTE: Subjects with plaque psoriasis can also be classified to have psoriatic arthritis (confirmed by CASPAR criteria [APPENDIX 13])
- b) For subjects with generalized pustular psoriasis:
  - i) Men and women with a prior history of or newly diagnosed generalized pustular psoriasis based on JDA criteria (APPENDIX 17)
  - ii) Have generalized pustular psoriasis and have been on a stable treatment regimen for at least 2 weeks prior to Day 1
  - iii) At Screening Visit and Day 1, have erythematous lesions with pustules involving ≥10% of body surface area (ie, score of at least 2 on this skin symptom [APPENDIX 17])
  - iv) At Screening Visit, total JDA severity index score <14 (APPENDIX 17)
  - v) Deemed by the investigator to be a candidate for phototherapy or systemic therapy
- c) For subjects with erythrodermic psoriasis:

- i) Men and women with a prior history of or newly diagnosed erythrodermic psoriasis
- ii) A history of plaque-type psoriasis
- iii) At Screening Visit and Day 1, have ≥80% of BSA involvement
- iv) Deemed by the investigator to be a candidate for phototherapy or systemic therapy

## 3) Age and Reproductive Status

- a) Men and women aged  $\geq 20$  years at the time of Screening Visit
- b) Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at Screening Visit, and a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of study drug
- c) Women must not be pregnant, lactating, breastfeeding, or planning pregnancy during the study period. Women must not enroll even if lactation or breastfeeding is interrupted.
- d) Women of childbearing potential must agree to use correctly a highly effective method(s) of contraception for the duration of treatment (52 weeks) with study drug(s) BMS-986165 plus 5 half-lives of study drug (3 days) plus 30 days (duration of ovulatory cycle) for a total of 33 days post-treatment completion (total of 33 days after last dose of study drug). WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements, but must still undergo pregnancy testing as described in this protocol
- e) Male subjects who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (APPENDIX 4) for the duration of treatment with study treatment(s) plus 5 half-lives of the study treatment (3 days) for a total of 3 days post-treatment completion. In addition, male subjects must be willing to refrain from sperm donation during this time

Investigators shall counsel WOCBP, and male subjects who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, (APPENDIX 4) which have a failure rate of < 1% when used consistently and correctly.

#### 5.2 Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

#### 1) Target Disease Exceptions

- a) Subjects with guttate, inverse, or drug-induced psoriasis at Screening or Day 1.
  - Note: the study allows men and women diagnosed with generalized pustular psoriasis or erythrodermic psoriasis.

#### 2) Infectious/Immune-related Exclusions

- a) History or evidence of outpatient active infection and/or febrile illness within 7 days of Day 1
- b) History of serious bacterial, fungal, or viral infections requiring hospitalization and/or intravenous (IV) antibiotic treatment within 60 days prior to Day 1
- c) Any untreated bacterial infection within 60 days prior to Day 1
- d) Any ongoing evidence of chronic, bacterial infection (eg chronic pyelonephritis, chronic osteomyelitis, chronic bronchiectasis)
- e) Any history of proven infection of a joint prosthesis in which the prosthesis was not removed or replaced, or received antibiotics for suspected infection of a joint prosthesis in which the prosthesis was not removed or replaced
- f) Received live vaccines within 60 days prior to Day 1, or plans to receive a live vaccine during the study, or within 60 days after completing study treatment
- g) Presence of herpes zoster lesions at Screening or Day 1
- h) History of serious herpes zoster or serious herpes simplex infection which includes, but is not limited to, any episode of disseminated herpes simplex, multidermatomal herpes zoster, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (recurrent is defined as 2 episodes within 2 years)
- i) Evidence of, or test positive for, hepatitis B virus (HBV) at Screening. Positive hepatitis B lab testing is defined as: 1) Positive hepatitis B surface antigen (HBsAg+) OR 2) Presence of HBV deoxyribonucleic acid (DNA) OR 3) Positive hepatitis B core antibody subjects with detectable HBV DNA by Polymerase Chain Reaction (PCR) OR 4) Positive hepatitis B surface antibody subjects with detectable HBV DNA by PCR.
  - Subjects with negative HBsAg but positive anti-HBs Ab, and/or positive anti-HBc Ab must also be tested for quantitative HBV DNA. Subjects with HBV DNA ≥2.1 Log copy/mL (20 IU/mL) are excluded from the study. Subjects with HBV DNA < 2.1 Log copy/mL (20 IU/mL) can be enrolled in the study but must undergo periodic monitoring of HBV DNA and liver enzymes, such as AST and ALT. Monitoring should be performed every 4 weeks throughout the duration of the study and at the Safety Follow-Up visit at Week 56.
- j) Evidence of, or test positive for, hepatitis C virus (HCV) at Screening. A positive test for HCV is defined as: 1) positive for hepatitis C antibody (anti-HCV Ab) **AND** 2) positive via a confirmatory test for HCV (eg, HCV PCR)
- k) Positive for human immunodeficiency virus by antibody testing (HIV-1 and -2 Ab) at Screening
- 1) Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the subject's immune status (eg, history of opportunistic infections [eg, *Pneumocystis jirovecii* pneumonia, histoplasmosis, or coccidioidomycosis], history of splenectomy, primary immunodeficiency)

#### 3) Any of the following TB criteria:

- a) History of active TB prior to Screening Visit, regardless of completion of adequate treatment
- b) Signs or symptoms of active TB (eg, fever, cough, night sweats, and weight loss) during Screening as judged by the investigator
- c) Any imaging of the chest (eg, chest x-ray, chest computed tomography [CT] scan) obtained during the Screening period or anytime within 6 months prior to Screening with documentation, showing evidence of current active or history of active pulmonary TB
- d) Latent TB infection (LTBI) defined as positive IFN gamma release assay (IGRA), by QuantiFERON®-TB Gold testing at Screening, in the absence of clinical manifestations

Note: Subject is eligible if (i) there are no current signs or symptoms of active TB AND (ii) subject has received adequate documented treatment for LTBI within 5 years of screening OR has initiated prophylactic treatment for LTBI per local guidelines and is rescreened after 1 month of treatment. To continue in the study, subject must agree to complete a locally-recommended course of treatment for LTBI.

Note: An IGRA test that is indeterminate with no signs or symptoms of active TB must be retested for confirmation. If the second test is again indeterminate, the subject will be excluded from the study. If the retest is positive, the subject should be treated as having LTBI. If the retest is negative, subject may be eligible provided no other exclusion criteria for TB are met.

## 4) Medical History and Concurrent Diseases

- a) Any major surgery within 8 weeks prior to Day 1, or any planned surgery for the first 52 weeks of the study
- b) Has donated blood >500 mL within 4 weeks prior to Day 1, or plans to donate blood during the course of the study
- c) Drug or alcohol abuse, as determined by the investigator, within 6 months prior to Day 1
- d) Medical marijuana or prescription marijuana taken for medicinal reasons
- e) Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, psychiatric, neurologic, immunologic, or local active infection/infectious illness) that, in the investigator's judgment or after consultation with the Medical Monitor, will substantially increase the risk to the subject if he or she participates in the study
- f) Unstable cardiovascular disease, defined as a recent clinical cardiovascular event (eg, unstable angina, myocardial infarction, stroke, rapid atrial fibrillation) in the last 3 months prior to Screening, or a cardiac hospitalization (eg, revascularization procedure, pacemaker implantation) within 3 months prior to Screening

- g) Has uncontrolled arterial hypertension characterized by a systolic blood pressure (BP) >160 mm Hg or diastolic BP >100 mm Hg
  - Note: Determined by 2 consecutive elevated readings. If an initial BP reading exceeds this limit, the BP may be repeated once after the subject has rested sitting for  $\geq 10$  minutes. If the repeat value is less than the criterion limits, the second value may be accepted
- h) Class III or IV congestive heart failure by New York Heart Association Criteria
- i) Has cancer or history of cancer (solid organ or hematologic including myelodysplastic syndrome) or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell or squamous cell carcinoma, or carcinoma of cervix in situ that has been treated with no evidence of recurrence)
- j) Any uncontrolled neuropsychiatric illness judged as clinically significant by the investigator during Screening or at Day 1

#### OR

Any lifetime history of suicidal ideation, suicidal behavior, or suicidal attempts by medical history or by electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) documentation, or by answering "yes" to Question 4 or 5 for suicidal ideation on the eC-SSRS at Screening or at Day 1, or is clinically deemed to have a suicide risk by the investigator

- k) Prior exposure to BMS-986165
- l) If the subject has received biologics previously, the following exclusion criteria for washout will apply:
  - i) Antibodies to IL-12, IL-17, or IL-23 (eg, ustekinumab, secukinumab, tildrakizumab, ixekizumab, or guselkumab) within 6 months of Day 1
  - ii) TNF inhibitor(s) (eg etanercept, adalimumab, infliximab, certolizumab) within 2 months of Day 1
  - iii) Agents that modulate integrin pathways to impact lymphocyte trafficking (eg natalizumab), or agents that modulate B cells or T cells (eg, alemtuzumab, abatacept, or visilizumab) within 3 months of Day 1
  - iv) Rituximab within 6 months of Day 1
- m) Has received systemic nonbiologic psoriasis medications and/or any systemic immunosuppressants (including, but not limited to, methotrexate [MTX], azathioprine, cyclosporine, JAK inhibitors, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus, oral or injectable corticosteroids, retinoids, 1,25-dihydroxy vitamin D3 and analogs, psoralens, sulfasalazine, or fumaric acid derivatives) within 4 weeks prior to Day 1 with the following exceptions:
  - i) For subjects with erythrodermic psoriasis or generalized pustular psoriasis, use of prednisone or its equivalent at a daily dose  $\leq 10$  mg/day is permitted

- ii) For subjects with generalized pustular psoriasis, one of the following agents is permitted: cyclosporine, methotrexate, or retinoids
- iii) For subjects with erythrodermic psoriasis, concomitant use of cyclosporine is permitted until Week 2
- n) Has used leflunomide within 6 months prior to Day 1
- o) Has used opioid analgesics within 4 weeks prior to Day 1
- p) Has received lithium, antimalarials, or intramuscular (IM) gold within 4 weeks of the first administration of any study medication
- q) Has received phototherapy (including either oral and topical PUVA light therapy, (UVB) or self-treatment with tanning beds or therapeutic sunbathing) within 4 weeks prior to Day 1
- r) Has used topical medications/treatments that could affect psoriasis evaluation (including, but not limited to, ultra-high to moderate potency corticosteroids (Classes I-V), >3% salicylic acid, urea, alpha- or beta-hydroxyl acids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, picrolimus, and tacrolimus) within 2 weeks prior to Day 1
  - Note: Low potency topical steroids (WHO Classes VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha- or beta- hydroxy acids or other ingredients which are pharmacologically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit.
- s) Use of shampoos that contain corticosteroids, coal tar, >3% salicylic acid, or vitamin D3 analogues within 2 weeks prior to Day 1
- t) Has received an experimental antibody or experimental biologic therapy within the previous 6 months, **OR** received any other experimental therapy or new investigational agent within 30 days or 5 half-lives (whichever is longer) prior to Day 1 **OR** is currently enrolled in an investigational study
- u) The following conditions for subjects with generalized pustular psoriasis:
  - i. Drug-induced generalized pustular psoriasis
  - ii. Subcorneal pustular dermatosis
  - iii. Previous psoriasis vulgaris who experienced temporary pustulation
  - iv. Circinate annular form of generalized pustular psoriasis
- v) For subjects with psoriatic arthritis:
  - i. Received any parenteral corticosteroid injections within 6 weeks of Screening
- w) Any other sound medical, psychiatric and/or social reason as determined by the investigator

#### 5) Physical and Laboratory Test Findings

- a) At Screening
  - i) Absolute WBC count <3000/mm<sup>3</sup>
  - ii) Absolute lymphocyte count <500/mm<sup>3</sup>
  - iii) Absolute neutrophil count <1000/mm<sup>3</sup>
  - iv) Platelet count <100,000/mm<sup>3</sup>
  - v) Hemoglobin <9 g/dL
  - vi) ALT and/or AST >3X upper limit of normal (ULN)
  - vii) Total, unconjugated, and/or conjugated bilirubin >2X ULN
  - viii) Thyroid-stimulating hormone (TSH) outside the normal reference range

**AND** 

Free T4 (thyroxine) or T3 (triiodothyronine) outside the normal reference range

- b) ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the subject if participating in the study
- c) Renal impairment based on an estimated glomerular filtration rate (eGFR) <45 mL/min
- d) Inability to be venipunctured and/or tolerate venous access
- e) Any other significant laboratory abnormalities that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study
- f)  $(1\rightarrow 3)$ -beta-D-glucan positive

#### 6) Allergies and Adverse Drug Reaction

a) History of any significant drug allergy (such as anaphylaxis)

## 7) Other Exclusion Criteria

- a) Prisoners or subjects who are involuntarily incarcerated. (Note: under certain specific circumstances a person who has been imprisoned may be included or permitted to continue as a subject. Strict conditions apply and BMS approval is required).
- b) Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
- c) Inability to comply with restrictions and prohibited activities/treatments as listed in the study protocol
- d) Site personnel or their immediate family

# 5.3 Lifestyle Restrictions

General skin care measures (with above restrictions for topical treatments) that are standard for subjects with plaque psoriasis are permitted. Subjects should avoid excessive sun exposure and avoid risks that are known to provoke flare of psoriasis.

## 5.3.1 Meals and Dietary Restrictions

Study treatment may be taken without regard to meals; however, subjects are required to fast for a minimum of 10 hours before visits on which fasting lipid samples will be drawn.

# 5.3.2 Caffeine, Alcohol and Tobacco

No restrictions are required; however extensive use of caffeine, alcohol, and tobacco should be avoided.

# 5.3.3 Activity

No restrictions are required; however, unusual physical exertion should be avoided during the study.

#### 5.4 Screen Failures

Screen failures are defined as subjects who consent to participate in the clinical study but are not subsequently enrolled in the study for any reason. A minimal set of screen failure information is required to ensure transparent reporting of screen failure subjects, to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements, and to respond to queries from regulatory authorities. Minimal set of screen failure information includes date of consent, demography, screen failure details (ie, eligibility criteria that the subject did not meet), and any SAEs during the Screening period.

# 5.4.1 Retesting During Screening or Rescreening

For laboratory parameters that initially do not meet eligibility requirements, a single retest within the 28-day screening period is permitted before subject is declared a screen failure. This is an effort to find all possible well-qualified subjects. Consultation with the Medical Monitor may be needed to identify whether repeat testing of any particular parameter would be clinically relevant.

The study permits the rescreening (after the end of the initial 28-day screening period) of a subject who discontinues the study as a pretreatment failure (ie, the subject fails to meet eligibility criteria and has not been treated). The subject must be reconsented, will be assigned a new identification number, and a full Screening Visit must be performed again. A subject can only be rescreened 1 time (ie, if the subject fails 1 rescreening attempt, no additional rescreening is allowed). Depending on the timing of rescreening, repeat chest imaging may not be required. Duration of existing treatments and required discontinuation periods shall be considered relative to the new Screening Visit and/or enrollment.

The most current result prior to enrollment is the value by which study inclusion will be assessed, as it represents the subject's most current clinical state.

#### 6 TREATMENT

Study treatment is defined as any investigational treatment(s), marketed product(s), placebo, or medical device intended to be administered to a study subject according to the study randomization or treatment allocation.

Study treatment includes both Investigational [Medicinal] Product (IP/IMP) and Non-investigational [Medicinal] Product (Non-IP/Non-IMP) and can consist of the following: BMS-986165.

An IP, also known as IMP in some regions, is defined as a pharmaceutical form of an active substance or placebo being tested or used as a reference in a clinical study, including products already with a marketing authorization but used or assembled (formulated or packaged) differently than the authorized form, or used for an unauthorized indication, or when used to gain further information about the authorized form.

Other medications used as support or escape medication for preventative, diagnostic, or therapeutic reasons, as components of the standard of care for a given diagnosis, may be considered as noninvestigational products. Table 4 shows the study treatments for Protocol IM011066.

Table 4: Study Treatments for Study Number

| Product Description/Class and Dosage Form | Potency | IP/Non-<br>IMP | Open-<br>Label | Packaging/Appearance | Storage<br>Conditions<br>(per label) |
|---|---|---|---|---|---|
| BMS-986165<br>tablet | 6 mg | IP | Open-<br>Label | Bottle | Store at 15 to<br>25°C; Store in a<br>tightly closed<br>container; Protect<br>from light |

#### 6.1 Treatments Administered

Study treatment will be administered as described in Section 4.1.2. The selection and timing of dose for each subject is in Table 5:

Table 5: Selection and Timing of Dose

| Study Treatment | Unit dose<br>strength(s)/Dosage<br>level(s) | Dosage formulation<br>Frequency of<br>Administration | Route of<br>Administration |
|---|---|---|---|
| 6 mg QD BMS-986165 | 6 mg | 1 active tablet QD in the morning | oral |

Abbreviations: QD = once daily

# **6.2** Method of Treatment Assignment

Before the study is initiated, each user (at investigative sites) will receive log-in information and directions on how to access the interactive response technology (IRT) system. At the time of the Screening Visit, immediately after informed consent is obtained and before any study-related procedures are performed, the investigative site will access the enrollment option of the IRT system for assignment of a subject number for all subjects including subjects not subsequently treated. The subject number is assigned sequentially by the system and will be unique across all sites. All enrolled subjects, including those not dosed, will be assigned sequential subject numbers. The subject number may not be used for any other subject. If a subject is rescreened, they will be given a new identification number.

A kit will contain adequate study treatment for a 4-week supply. At subsequent visits, when new treatment kits need to be provided, the investigative site will access the IRT to obtain the kit number to assign to the subject. Study treatment will be dispensed at study visits as shown in the Schedule of Activities (Section 1.2).

#### 6.3 Blinding

This is an open-label study, blinding procedures are not applicable.

## 6.4 Dosage Modification

There is no provision for dose modification of study treatment. If a subject interrupts treatment due to an AE, study treatment can be restarted in consultation with the Medical Monitor.

# 6.5 Preparation/Handling/Storage/Accountability

The IP should be stored in a secure area according to local regulations. It is the responsibility of the investigator to ensure that IP is only dispensed to study subjects. The IP must be dispensed only from official study sites by authorized personnel according to local regulations.

The product storage manager should ensure that the study treatment is stored in accordance with the environmental conditions (temperature, light, and humidity) as determined by BMS. If concerns regarding the quality or appearance of the study treatment arise, the study treatment should not be dispensed and BMS should be contacted immediately.

Investigational product documentation (whether supplied by BMS or not) must be maintained, that includes all processes required to ensure drug is accurately administered. This includes documentation of drug storage, administration and, as applicable, storage temperatures, reconstitution, and use of required processes (eg, required diluents, administration sets).

Guidance and information for final disposition of unused study treatment are provided in APPENDIX 2.

#### 6.5.1 Retained Samples for Bioavailability/Bioequivalence

Not applicable.

#### 6.6 Treatment Compliance

Study treatment compliance will be periodically monitored using standard drug accountability procedures (comparing the number of tablets returned to number dispensed, considering the expected regimen and any reported missed doses). Drug accountability will be reviewed by the investigative site staff at each visit to confirm treatment compliance. Site staff will discuss any discrepancies with the subject and remind the subject of the importance of compliance with the assigned regimen. A real-time monitoring platform may be used.

# 6.7 Concomitant Therapy

#### 6.7.1 Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications during the study are described below. Medications taken within 4 weeks prior to study drug administration must be recorded on the CRF.

- 1) Exposure to any investigational drug or placebo outside of the current study
- 2) Use of any medications/therapy that would aggravate psoriasis. These include agents such as lithium, antimalarials (quinacrine, chloroquine, and hydroxychloroquine), propranolol, indomethacin, and quinidine unless it is considered necessary for the subject's welfare and/or treatment of an AE/SAE.
- 3) Use of opioid analgesics unless it is considered necessary for the subject's welfare and/or treatment of an AE/SAE
- 4) Phototherapy, use of tanning booths or therapeutic sunbathing
- 5) Any use of biologic medications (eg, adalimumab, etanercept, infliximab, ustekinumab)
- 6) Any use of oral psoriasis medications (eg, methotrexate, cyclosporine, retinoids, fumaric acid derivatives) for any indication
  - a. For subjects with generalized pustular psoriasis, one of the following agents is permitted: cyclosporine, methotrexate, or retinoids.
  - b. For subjects with erythrodermic psoriasis, concomitant use of cyclosporine is permitted until Week 2.
- 7) Any use of oral or injectable corticosteroids (eg, prednisone, methylprednisolone), unless it is considered necessary for the subject's welfare and/or treatment of an AE/SAE
  - a. For subjects with erythrodermic psoriasis or generalized pustular psoriasis, use of prednisone or its equivalent at a daily dose  $\leq$  10 mg/day is permitted.
  - b. Otic, ophthalmic, nasal, or inhaled corticosteroids within recommended doses and with no systemic effects are permitted.
- 8) Any topical medications/treatments, which are used for any indication, that could affect psoriasis evaluation (including, but not limited to, ultra-high to moderate potency corticosteroids (WHO Classes I-V), >3% salicylic acid, urea, alpha- or beta-hydroxyl acids,

anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, picrolimus, and tacrolimus).

Exception: The following topical treatments may be initiated only at Week 24 per investigator's discretion in subjects who have (See Section 4.1.4):

• Ultra-high to moderate potency corticosteroids (Classes I-V), >3% salicylic acid, urea, alpha- or beta- hydroxyl acids, anthralin, calcipotriene, vitamin D derivatives, retinoids, tazarotene

Note: Low potency topical steroids (WHO Classes VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha- or beta-hydroxy acids or other ingredients which are pharmacologically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit.

9) Any medicated shampoos that contain corticosteroids, coal tar, >3% salicylic acid, or vitamin D3 analogues

Exception: The above shampoos may be initiated only at Week 24 per investigator's discretion in subjects who have (See Section 4.1.5).

## 10) Live vaccination

No concomitant medications (prescription, over-the-counter or herbal) are to be administered during study unless they are prescribed for treatment of specific clinical events. Any concomitant therapies must be recorded on the CRF.

The investigator should contact and confirm agreement with the Medical Monitor prior to the administration of any concomitant medications.

#### 6.7.2 Permitted Concomitant Medications

Stable doses of concomitant medication for chronic medical conditions are permitted as long as neither the medication nor the medical condition meet exclusion criteria as detailed in Section 5.2. Dose adjustments of these medications should be avoided during the study unless clinically indicated. If a dose adjustment of these medications should occur, they must be recorded on the Concomitant Medications electronic case report form (eCRF) or the Procedures and Significant nondrug therapies eCRF. The investigator should instruct the subject to notify the study site about any new treatments he/she takes after the start of the study treatment. All medications and significant nondrug therapies (including physical therapy and blood transfusions) administered after the subject starts study treatment must be listed on the Concomitant Medications eCRF or the Procedures and Significant non-drug therapies eCRF.

#### Note:

• Low potency topical steroids (WHO Class VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha- or beta-hydroxy acids or

other ingredients which are pharmacologically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit.

- For subjects with erythrodermic psoriasis or generalized pustular psoriasis, use of prednisone or its equivalent at a daily dose ≤ 10 mg/day is permitted.
- For subjects with erythrodermic psoriasis, concomitant use of cyclosporine is permitted until Week 2.
- For subjects with generalized pustular psoriasis, one of the following agents is permitted: cyclosporine, methotrexate, or retinoids.

#### 6.7.3 Rescue Medications

At Week 24, a subject who has an may be treated with restricted topicals or shampoos, respectively, as described in Section 6.7.1 at the investigator's discretion. These treatments may only be initiated at Week 24, and not at subsequent time points. A subject who is initiated on these treatments at Week 24 may use them as needed per the investigator's judgment through Week 52.

# 6.8 Treatment After the End of the Study

At the end of the study, the investigator should ensure that subjects continue to receive appropriate standard of care to treat the condition under study.

In addition, for subjects who continue to demonstrate clinical benefit, BMS may continue to provide study treatment via a rollover extension study requiring approval by responsible health authority and ethics committee, or through another mechanism at the discretion of BMS.

BMS reserves the right to terminate access to BMS supplied study treatment if any of the following occur: a) the study is terminated due to safety concerns; b) the development of BMS-986165 is terminated for other reasons, including but not limited to lack of efficacy and/or not meeting the study objectives; c) the subject can obtain medication from a government sponsored or private health program. In all cases BMS will follow local regulations.

#### 7 DISCONTINUATION CRITERIA

# 7.1 Discontinuation from Study Treatment

Subjects MUST discontinue IP (and non-IP at the discretion of the investigator) for any of the following reasons:

- Subject requests to stop study treatment. Subjects who discontinue study treatment early should remain in the study for protocol-specified procedures. The only exception to this is when a subject specifically withdraws consent for any further contact with him/her or persons previously authorized by subject to provide this information.
- Any clinically significant AE, laboratory abnormality, or intercurrent illness which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the subject. If treatment is discontinued due to an AE, the AE eCRF must be completed to show that the AE caused discontinuation.

- eGFR <45 mL/min on repeat assessment within 7 days
- Abnormal liver tests suggestive of drug-induced liver injury (DILI), as defined in Section 8.2.8 or if the investigator believes that it is in the best interest of the subject
- Subject reports suicidal ideation, suicidal behavior, or suicide attempts at any time after enrollment, or documents suicidal ideation by answering "Yes" to Question 4 or 5 on the eC-SSRS, or documents suicidal behavior on the eC-SSRS at any time during the study. The subject should then be immediately referred to a mental health professional for evaluation of suicide risk.
- The subject develops a malignancy, with the exception of a subject who develops non-melanoma skin cancer who may continue in the study at the discretion of the investigator
- Pregnancy, positive pregnancy test or subject expresses an interest in becoming pregnant (refer to Section 8.2.6)
- Subject develops active TB during the study or prematurely discontinues treatment for LTBI, or subject is noncompliant with LTBI therapy (refer to Section 8.4.4)
- Termination of the study or program by BMS
- Inability or failure to comply with protocol requirements in the opinion of the investigator
- Loss of ability to freely provide consent through imprisonment or involuntary incarceration for treatment of either a psychiatric or physical (eg, infectious disease) illness
- Subjects with a positive HBsAb at screening or a positive HBcAb at screening and negative HBV DNA (< 2.1 Log copy/mL [20 IU/mL] at screening have a quantitative HBV DNA ≥2.1 Log copy/mL (20 IU/mL) during study treatment

Refer to the Schedule of Activities (Section 1.2) for data to be collected at the time of treatment discontinuation and follow-up and for any further evaluations that can be completed.

All subjects who discontinue BMS-986165 should comply with protocol-specified follow-up procedures as outlined in Section 1.2. The only exception to this requirement is when a subject withdraws consent for all study procedures including post-treatment study follow-up or loses the ability to consent freely (ie, is imprisoned or involuntarily incarcerated for the treatment of either a psychiatric or physical illness). Replacement of subjects is not permitted.

If study treatment is discontinued prior to the subject's completion of the study, the reason for the discontinuation must be documented in the subject's medical records and entered on the appropriate eCRF page.

#### 7.1.1 Temporary Discontinuation

Temporary study treatment discontinuation is only allowed if the subject develops an AE which, in the opinion of the investigator, indicates that it is in the subject's best interest that the study

treatment be placed on hold. Study treatment in this situation should be stopped until the AE is medically treated and/or has resolved per investigator judgment.

Any temporary study treatment discontinuation as well as restart must be documented on the corresponding eCRF.

# 7.1.2 Post-Study Treatment Follow-Up

Post-study follow-up is of critical importance and is essential to preserving subject safety and the integrity of the study. Subjects who discontinue study treatment must continue to be followed for collection of outcomes and/or survival follow-up data as required and in line with Section 4 until death or the conclusion of the study.

Subjects who discontinue study treatment should be encouraged to undergo all study-related visits for the full treatment period in order to support the final efficacy and safety analysis.

## 7.2 Discontinuation from the Study

Subjects who request to discontinue study treatment will remain in the study and must continue to be followed for protocol-specified follow-up procedures as specified in Section 1.2. The only exception to this is when a subject specifically withdraws consent for any further contact with him/her or persons previously authorized by subject to provide this information.

- Subjects should notify the investigator of the decision to withdraw consent from future follow-up in writing, whenever possible.
- The withdrawal of consent should be explained in detail in the medical records by the investigator and entered on the appropriate CRF page.
- In the event that vital status (whether the subject is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.
- If the subject withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.

# 7.3 Lost to Follow-up

- All reasonable efforts must be made to locate subjects to determine and report their ongoing status. This includes follow-up with persons authorized by the subject.
- Lost to follow-up is defined by the inability to reach the subject after a minimum of **three** documented phone calls, faxes, or emails as well as lack of response by subject to one registered mail letter. All attempts should be documented in the subject's medical records.
- If it is determined that the subject has died, the site will use permissible local methods to obtain date and cause of death.
- If investigator's use of third-party representative to assist in the follow-up portion of the study has been included in the subject's informed consent, then the investigator may use a Sponsor retained third-party representative to assist site staff with obtaining subject's

contact information or other public vital status data necessary to complete the follow-up portion of the study.

- The site staff and representative will consult publicly available sources, such as public health registries and databases, in order to obtain updated contact information.
- If after all attempts, the subject remains lost to follow-up, then the last known alive date as
  determined by the investigator should be reported and documented in the subject's medical
  records.

#### 8 STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and timing are summarized in the Schedule of Activities (Section 1.2) and described in Section 4.1.
- Protocol waivers or exemptions are not allowed.
- All significant safety concerns must be discussed with the Medical Monitor immediately
  upon occurrence or awareness to determine if the subject should continue or discontinue
  treatment.
- Adherence to the study design requirements, including those specified in the Schedule of Activities (Section 1.2), is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential subjects meet all eligibility criteria before enrollment. Enrollment should not occur until at least 8 days after the Screening Visit

   The investigator will maintain a screening log to record details of all subjects screened and to confirm eligibility or record reasons for screening failure, as applicable.
- Procedures conducted as part of the subject's routine clinical management (eg, blood count) and obtained before signing of informed consent may be utilized for screening or baseline purposes provided the procedure meets the protocol-defined criteria and has been performed within the timeframe defined in the Schedule of Activities (Section 1.2).
- For several assessments, appropriate training will be provided to investigators and designated personnel at sites. Only those individuals trained and certified to perform these assessments will be performing them during the study.

#### 8.1 Efficacy Assessments

Every effort must be made to ensure that the same evaluator(s) complete the investigator-administered assessments for each subject at each visit. If the evaluator(s) is unable to complete the evaluation, then a qualified individual with overlapping experience may perform the evaluation. Documentation of who performed the evaluation is to be recorded in source documents. Assessments are to be performed at approximately the same time of day throughout the duration of the study.

Baseline assessments must be performed per protocol. Procedures not specified in the protocol that are part of standard care may be performed if they do not interfere with study procedures; any data arising from such procedures are not to be reported in the eCRF.

# 8.1.1 Investigator-administered Assessments

# 8.1.1.1 static Physician Global Assessment (sPGA)

The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). sPGA assessments should be performed by a trained physician (eg, dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients. Every effort should be made to ensure that the physician or designee who performed the sPGA evaluations for a subject at enrollment performs the sPGA for that subject at all subsequent visits (see APPENDIX 5).

## 8.1.1.2 Psoriasis Area and Severity Index (PASI)

The PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. The PASI can also be used to assess response to treatment. The PASI 50 is the proportion of subjects who experience at least a 50% improvement in PASI score as compared with the baseline value. The PASI 75 are defined similarly. BMS will host a training session prior to initiation of the study to demonstrate proper PASI scoring. All PASI assessments should be performed by a trained physician (dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients (see APPENDIX 6).

# 8.1.1.3 Body Surface Area (BSA)

Measurement of psoriasis BSA involvement is estimated using the handprint method with the size of a subject's handprint (including fingers and thumb) representing 1% of BSA involved. The total BSA = 100% with breakdown by body region as follows: head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), trunk including axillae and groin = 30% (30 handprints), lower extremities including buttocks = 40% (40 handprints). BSA assessments should be performed by a dermatologist or appropriately trained investigator who is experienced in the assessment of psoriasis patients.







# 8.1.1.12 Severity Criteria for Generalized Pustular Psoriasis by the Japanese Dermatological Association (JDA)

The severity will be categorized as: mild (0 to 6), moderate (7 to 10) or severe (11 to 17) by total score. Total score (0 to 17) will be calculated by the evaluation of skin symptoms (0 to 9) and systemic symptoms and laboratory findings (0 to 8) (see APPENDIX 17).

# 8.1.2 Subject-Reported Assessments





# 8.1.2.6 Psoriatic Arthritis Screening and Evaluation (PASE) Questionnaire

The PASE questionnaire will be administered at screening in subjects with psoriatic arthritis type complaints. The PASE questionnaire is a self-administered tool that is used to screen for psoriatic arthritis among subjects who have psoriasis. The PASE questionnaire consists of 15 questions subdivided into 7 questions focusing on symptoms of psoriatic arthritis, and 8 questions focusing on the impact of psoriatic arthritis on function. Each question is scored on a 1 to 5 scale, with a maximum score of 75. A score of 47 or above has been shown to distinguish between psoriatic arthritis and non-psoriatic arthritis. This questionnaire is only intended to be a screening tool for psoriatic arthritis and does not replace a comprehensive musculoskeletal exam performed by a rheumatologist. The PASE questionnaire should take 6 to 10 minutes to complete and is only done at Screening (See APPENDIX 23).

#### 8.2 Adverse Events

The definitions of an AE or SAE can be found in APPENDIX 3.

AEs will be reported by the subject (or, when appropriate, by a caregiver, surrogate, or the subject's legally authorized representative).

The investigator and any designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study treatment or the study, or that caused the subject to discontinue before completing the study.

**Contacts for SAE reporting are specified in APPENDIX 3.** 

#### 8.2.1 Adverse Events of Interest

Adverse events of interest (AEIs) are AEs for a particular product or class of products that a Sponsor may wish to monitor carefully. Adverse events of interest may be serious or non-serious. Such events may require further investigation to better characterize and understand them. In the BMS-986165 clinical development program, certain skin-related AEs (eg, acne), infection AEs,

and CK elevation have been identified as potential AEIs; however, there has been no definitive assessment on the causal relationship between these events and treatment with BMS-986165. Additionally, given a potential association between treatment for autoimmune diseases and increased risk for cancer, malignancy has been identified as a potential AEI. Suicidal ideation/behavior and an increased risk of cardiovascular disease may also be prevalent in patients with psoriasis. Therefore, additional information about certain skin-related AEs, infection AEs, CK elevation, suicidal ideation/behavior, cardiovascular events, and malignancy may be collected on the CRF in order to better characterize and understand them.

# 8.2.2 Time Period and Frequency for Collecting AE and SAE Information

The collection of non-serious AE information should begin at initiation of study treatment until discharge from the study (ie, final study visit for a given subject), at the timepoints specified in the Schedule of Activities (Section 1.2).

The Reference Safety Information in sections 5.6.1 and 5.6.2 of the IB should be used to determine expectedness of SAEs for expedited reporting. Following the subject's written consent to participate in the study, all SAEs, whether related or not related to study drug, must be collected, including those thought to be associated with protocol-specified procedures.

All SAEs must be collected from the date of subject's written consent until 30 days after the final dose of the study drug or subject's participation in the study if the last scheduled visit occurs at a later time. Monitoring for SAEs will occur at every study visit.

- The investigator must report any SAE that occurs after these time periods and that is believed to be related to study drug or protocol-specified procedure. Medical occurrences that begin before the start of study treatment but after obtaining informed consent will be recorded on the appropriate section of the CRF.
- All SAEs will be recorded and reported to Sponsor or designee within 24 hours, as indicated in APPENDIX 3.
- The investigator will submit any updated SAE data to the Sponsor within 24 hours of this being available.

Investigators are not obligated to actively seek AEs or SAEs in former study subjects. However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he/she considers the event reasonably related to the study treatment or study participation, the investigator must promptly notify the Sponsor.

The method of evaluating and assessing causality of AEs and SAEs and the procedures for completing and reporting/transmitting SAE reports are provided in APPENDIX 3.

# 8.2.3 Method of Detecting AEs and SAEs

Adverse events can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a subject. (In order to prevent reporting bias, subjects should not be questioned regarding the specific occurrence of one or more AEs.)

#### 8.2.4 Follow-up of AEs and SAEs

- Non-serious AEs should be followed to resolution or stabilization, or reported as SAEs if they become serious (see APPENDIX 3).
- Follow-up is also required for non-serious AEs that cause interruption or discontinuation of study treatment and for those present at the end of study treatment as appropriate.
- All identified non-serious AEs must be recorded and described on the non-serious AE page of the CRF. Completion of supplemental CRFs may be requested for AEs and/or laboratory abnormalities that are reported/identified during the course of the study.

After the initial AE/SAE report, the investigator is required to proactively follow each subject at subsequent visits/contacts. All SAEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the subject is lost to follow-up (as defined in Section 7.3).

Further information on follow-up procedures is given in APPENDIX 3.

## 8.2.5 Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the Sponsor of SAEs is essential so that legal obligations and ethical responsibilities toward the safety of subjects and the safety of a product under clinical investigation are met.
- An investigator who receives an investigator safety report describing SAEs or other specific safety information (eg, summary or listing of SAEs) from the Sponsor will file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

Sponsor or designee will be reporting AEs to regulatory authorities and ethics committees according to local applicable laws including European Directive 2001/20/EC and Food and Drug Administration (FDA) Code of Federal Regulations 21 CFR Parts 312 and 320. A SUSAR (Suspected, Unexpected Serious Adverse Reaction) is a subset of SAEs and will be reported to the appropriate regulatory authorities and investigators following local and global guidelines and requirements.

# 8.2.6 Pregnancy

In the event a subject becomes pregnant during the trial, the study treatment must be discontinued immediately. If the subject becomes pregnant while on treatment or within 3 days of discontinuing study treatment, the investigator must immediately notify Drug Safety of this event and complete and forward a Pregnancy Surveillance Form to Drug Safety within 24 hours of awareness of the event and in accordance with SAE reporting procedures described in APPENDIX 3. The investigator must also notify the Medical Monitor or designee of this event within 24 hours of awareness of pregnancy.

The pregnant subject will need to be followed up until the conclusion of the pregnancy for pregnancy outcomes. The safety data of the subject will continue to be collected under the same rules as instructed in Section 7.1.

Any pregnancy that occurs in a female partner of a male study subject should be reported to Drug Safety. In order for Sponsor or designee to collect any pregnancy surveillance information from the female partner, the female partner must sign an ICF for disclosure of this information. Information on this pregnancy will be collected on the Pregnancy Surveillance Form.

#### 8.2.7 Laboratory Test Result Abnormalities

The following laboratory test result abnormalities should be captured on the AE eCRF page.

- Any laboratory test result that is clinically significant or meets the definition of an AE or SAE
- Any laboratory test result abnormality that required the subject to have study treatment discontinued or interrupted
- Any laboratory test result abnormality that required the subject to receive specific corrective therapy

If a laboratory test result meets the definition of an AE or SAE, the laboratory test result should be reported as an AE or SAE and submitted to Drug Safety, as specified in APPENDIX 3.

It is expected that wherever possible, the clinical rather than laboratory term would be used by the reporting investigator (eg, anemia versus low hemoglobin value).

## 8.2.8 Potential Drug-Induced Liver Injury (DILI)

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 8.2 and APPENDIX 3 for reporting details). Wherever possible, timely confirmation of initial liver-related laboratory abnormalities should occur prior to the reporting of a potential DILI event.

Potential DILI is defined as:

1) ALT or AST elevation > 3 times ULN

#### **AND**

2) Total bilirubin > 2 times ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase),

#### **AND**

3) No other immediately apparent possible causes of liver function test elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, preexisting chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic.

# 8.2.9 Other Safety Considerations

Any significant worsening of a preexisting medical condition noted during interim or final physical examinations, ECG, x-ray filming, any other potential safety assessment required or not required by protocol should also be recorded as a non-serious or serious AE, as appropriate, and reported accordingly.

#### 8.3 Overdose

For this study, taking more than 2 days' study medication within a 24-hour time period will be considered an overdose.

In the event of an overdose the investigator should:

- 1) Contact the Medical Monitor immediately
- 2) Closely monitor the subject for AEs/SAEs and laboratory abnormalities

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the Medical Monitor based on the clinical evaluation of the subject.

#### 8.4 Safety

Planned time points for all safety assessments are listed in the Schedule of Activities (Section 1.2).

## 8.4.1 Physical Examinations

A complete physical examination will include general appearance, vital signs, eyes, ears, nose, mouth, throat, neck, respiratory, cardiovascular, respiratory, GI/abdomen, lymphatic, musculoskeletal, skin, psychiatric and neurologic exams. A targeted physical examination will include any organ system associated with an AE or a laboratory abnormality.

#### 8.4.2 Vital Signs

Refer to Schedule of Activities (Section 1.2).

# 8.4.3 Electrocardiograms

A 12-lead ECG will be performed at the visits indicated in the Schedule of Activities (Section 1.2). The subject will remain supine for 5 to 10 minutes prior to the ECG, and must have their lab work done after the tracing so that the ECG results remain as accurate as possible. The ECG results will be read by the primary study investigator or a designee.

# 8.4.4 Tuberculosis Screening and Chest Imaging

Chest imaging results and PE are part of the process to assess a subject's eligibility, as outlined in Section 1.2 and as defined in exclusion criterion 3.c). Chest imaging (eg, chest x-ray, chest CT scan) at the Screening Visit is required if not already performed and documented within 6 months of obtaining written informed consent. A subject must not have active signs or symptoms of TB, as judged by the investigator, to be eligible for the study.

In addition to a complete PE and medical history to evaluate exposure to TB, all subjects will have a screening test, an IGRA (eg, QuantiFERON®-TB Gold) performed centrally. If unable to obtain central laboratory results, an IGRA test could be obtained locally, after consultation with the Medical Monitor. A subject with an indeterminate IGRA test result must be retested for confirmation. If the second result is again indeterminate, the subject will be excluded from the study. If the second result is positive, the subject should be considered as having LTBI provided there are no signs or symptoms of active TB. If the second result is negative, the subject may be eligible provided no other exclusion criterion for TB is met.

# 8.4.5 Clinical Safety Laboratory Assessments

Investigators must document their review of each laboratory safety report.

| Hem | atol | logy |
|-----|------|------|
|-----|------|------|

Hemoglobin (Hgb)

Hematocrit (Hct)

White Blood Cell Count, including differential

Platelet Count

#### Chemistry

Aspartate Aminotransferase (AST) Alanine Aminotransferase (ALT)

Total Bilirubin

Direct Bilirubin (if total bilirubin > ULN)

Alkaline Phosphatase

Lactate Dehydrogenase (LDH)

Creatinine

Blood Urea Nitrogen (BUN)

Uric Acid

Glucose (fasting at some visits)

Total Protein Albumin Sodium Potassium

Chloride Calcium Phosphorus

Creatine Phosphokinase (CK)\*

Estimated Glomerular Filtration Rate (eGFR)

#### Urinalysis

Protein

Glucose

Blood

Leukocyte Esterase

Specific Gravity

рН

Microscopic Examination (reflex if abnormal)

#### **Lipid Panel**

Cholesterol (total)

High Density Lipoprotein (HDL)

Low Density Lipoprotein (LDL)

Triglycerides

#### **Infectious Serologies**

Hepatitis C Antibody with reflex to Hepatitis C RNA if positive

Hepatitis B Surface Antigen (HBsAg)

Hepatitis B Surface Antibody (HBsAb)

Hepatitis B Core Antibody (HBcAb)

Hepatitis B DNA Viral Load (HBV DNA) \*\*

HIV-1 and -2 antibody

#### Other Analyses

Pregnancy test (WOCBP only: serum hCG test at screening, followed by urine hCG test every 4 weeks)

Follicle-Stimulating Hormone (FSH) (to confirm menopausal status [see APPENDIX 4], at screening)

Hemoglobin A1C

Thyroid-Stimulating Hormone (TSH)

If TSH above normal reference range, test free T4; if TSH below normal range, test free T4 & T3

Serum Immunoglobulin Levels (IgM, IgG, IgA, IgE)

 $(1\rightarrow 3)$ -beta-D glucan (at screening only)

<sup>\*</sup>If CK > 2.5X ULN, then reflex testing (ie, CK-MB, Troponin I will be required)

\*\*Testing for HBV DNA will occur every 4 weeks for subjects who are negative HBsAg but positive HBsAb and/or positive HBcAb with Hepatitis B virus DNA <2.1 log copies/mL [20IU/mL] at screening.

# 8.4.5.1 Estimated Glomerular Filtration Rate (eGFR)

Glomerular filtration rate will be estimated using the Modification of Diet in Renal Disease (MDRD) equation at screening.

The MDRD equation is as follows:<sup>45</sup>

eGFR = 
$$175 \times \text{standardized SCr}^{-1.154} \times \text{age}^{-0.203} \times 1.212$$
 [if black] or 0.742 [if female]

Note: GFR is expressed as mL/min/1.73 m<sup>2</sup> of body surface area and SCr (serum creatinine) is expressed in mg/dL.

Subjects with an eGFR <45 mL/min will be excluded from participation

## 8.4.6 Depression Monitoring

Depression will be monitored by administration of the eight-item Patient Health Questionnaire (PHQ-8) at Screening and during visits as outlined in Section 1.2.

#### 8.4.6.1 Eight-Item Patient Health Questionnaire (PHQ-8)

The PHQ-8 is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies. <sup>46</sup> Each of the 8 questions is based on a 2-week recall and scored on a scale of 0 to 3 by a tick box as: Not at All, Several Days, More than Half the Days, and Nearly Every Day. A score of  $\geq$ 10 is suggestive of moderate depressive symptoms (APPENDIX 24). <sup>47</sup> If a subject scores  $\geq$  15 on the PHQ-8 during the study, the investigator will review the situation and refer the subject to a mental health professional if deemed necessary.

## 8.4.7 Suicidal Ideation and Behavior Monitoring

Subjects in this clinical trial will be monitored for SIB by the eC-SSRS (Section 8.4.7.1) at the visits outlined in the Schedule of Activities (Section 1.2). Subjects who answer yes to questions 4 or 5 which indicates a suicidal ideation severity level of 4 or 5 or document suicidal behavior or suicidal attempts on the eC-SSRS will have their treatments discontinued and be immediately referred to a mental health professional for further evaluation. In addition, family members or caregivers of the subjects will be instructed to immediately report any suicidal ideation, suicidal behavior, or suicide attempt to the investigator.

## 8.4.7.1 electronic Columbia-Suicide Severity Rating Scale (eC-SSRS)

The eC-SSRS is a computer-automated, patient reported version of the C-SSRS instrument that defines 11 categories of SIB events. 48-50 The categories are as follows:

- Suicidal ideation
  - 1. Passive
  - 2. Active: Nonspecific (no method, intent, or plan)
  - 3. Active: Method, but no intent or plan
  - 4. Active: Method and intent, but no plan
  - 5. Active: Method, intent, and plan
- Suicidal behavior

- 1. Completed suicide
- 2. Suicide attempt
- 3. Interrupted attempt
- 4. Aborted attempt
- 5. Preparatory actions toward imminent suicidal behaviors
- Self-injurious behavior, no suicidal intent

Definitions of these categories can be found in APPENDIX 25.51










# 8.8 Health Economics OR Medical Resource Utilization and Health Economics

Health Economics/Medical Resource Utilization and Health Economics parameters will not be evaluated in this study.

## 9 STATISTICAL CONSIDERATIONS



# 9.2 Populations for Analyses

For purposes of analysis, the following analysis sets will be used in this trial:

**Enrolled Population:** All subjects who sign informed consent.

**As-treated Population:** All enrolled subjects who took at least one dose of study treatment.

**Plaque Psoriasis (PP) Population:** Subgroup of the As-treated population with plaque psoriasis per the inclusion criteria.

Generalized Pustular Psoriasis (GPP) Population: Subgroup of the As-treated population with generalized pustular psoriasis per the inclusion criteria.

Erythrodermic Psoriasis (EP) Population: Subgroup of the As-treated population with erythrodermic psoriasis per the inclusion criteria.



# 9.3 Endpoints

# 9.3.1 Primary Endpoints

- sPGA 0/1 response assessed as a proportion of subjects with a sPGA score of 0 or 1 at Week 16
- PASI 75 response assessed as a proportion of subjects who achieve a 75% improvement from baseline in the PASI score at Week 16







## 9.4 Efficacy Analyses

As this is a single-arm study, no statistical tests for treatment comparisons will be conducted. Categorical data will be summarized as frequency counts and percentages. Continuous data will be summarized using n, mean, standard deviation, median, minimum, and maximum unless otherwise specified. Efficacy variables will be summarized for all visits in which the variable is assessed. Complete details of the planned analyses will be documented in the statistical analysis plan and finalized before database lock. Summaries will be provided for plaque psoriasis (including psoriatic arthritis), generalized pustular psoriasis, and erythrodermic psoriasis subjects separately.

# 9.5 Safety Analyses

Safety data will be analyzed for AEs, SAEs, laboratory analytes, vital signs, ECGs, and suicidality and depression. Safety will be summarized using the As-treated population. Categorical data will be summarized as frequency counts and percentages. Continuous data will be summarized using n, mean, standard deviation, median, minimum, and maximum unless otherwise specified.

Additionally, safety data from the IM011-046 Japan subgroup will be integrated with safety data from IM011066 for descriptive summaries. Full details will be provided in the statistical analysis plan.

#### 9.5.1 Adverse Events

Treatment-emergent adverse events (TEAEs), SAEs and deaths, AEs leading to study treatment discontinuation, AEs by maximum severity, and AEs by relationship will be summarized by the MedDRA system organ class and preferred term. All TEAEs as well as each AE-adjudicated category (ie, infections, cardiovascular, and SIB) will also be summarized by preferred term sorted by decreasing frequency.

## 9.5.2 Vital Signs and ECGs

Vital signs and ECGs will be summarized as raw, change from baseline, and change from maximum postbaseline value. Incidence of abnormal ECG findings will also be summarized.

## 9.5.3 Clinical Laboratory Tests

Laboratory analytes will be summarized as raw, change from baseline, and change from maximum postbaseline value. Incidence of abnormal, high, or low values will be summarized.

## 9.5.4 Suicidality and Depression Assessments

Suicidality and depression will be assessed using eC-SSRS and PHQ-8. Data will be summarized, as applicable.

## 9.6 Other Analyses

## 9.6.1 Demographics and Baseline Data

Demographics and baseline data will be summarized using the As-treated population. Categorical data will be summarized as frequency counts and percentages. Continuous data will be summarized using n, mean, standard deviation, median, minimum, and maximum unless otherwise specified.

## 9.6.2 Prior and Concomitant Medications

Prior and concomitant medications, categorized by medication group and subgroup according to the WHO Drug Dictionary, will be summarized for the As-treated population. Medications with an end date prior to the first dose of study drug will be considered prior medications.



# 9.7 Interim Analysis

No interim analysis is currently planned.

## 10 REFERENCES

- 1. Fujita H, Terui T, Hayama K, et al. Japanese guidelines for the management and treatment of generalized pustular psoriasis: The new pathogenesis and treatment of GPP. J Dermatol 2018;45(11):1235-70.
- 2. Parisi R, Symmons DP, Griffiths CE, et al. Global epidemiology of psoriasis: a systematic review of incidence and prevalence. J Invest Dermatol 2013;133(2):377-85.
- 3. Kupetsky EA, Keller M. Psoriasis vulgaris: an evidence-based guide for primary care. J Am Board Fam Med 2013;26(6):787-801.
- 4. Global Report on Psoriasis. World Health Organization. Published 2016.
- 5. Langley RG, Krueger GG, Griffiths CE. Psoriasis: epidemiology, clinical features, and quality of life. Ann Rheum Dis 2005;64 Suppl 2:ii18-23; discussion ii4-5.
- 6. Queiro R, Tejon P, Alonso S, et al. Age at disease onset: a key factor for understanding psoriatic disease. Rheumatology (Oxford) 2014;53(7):1178-85.
- 7. Mrowietz U, Kragballe K, Reich K, et al. Definition of treatment goals for moderate to severe psoriasis: a European consensus. Arch Dermatol Res 2011;303(1):1-10.
- 8. Nestle FO, Kaplan DH, Barker J. Psoriasis. N Engl J Med 2009;361(5):496-509.
- 9. Mehta NN, Azfar RS, Shin DB, et al. Patients with severe psoriasis are at increased risk of cardiovascular mortality: cohort study using the General Practice Research Database. Eur Heart J 2010;31(8):1000-6.
- 10. Rheumatrex (methotrexate) [USPI]. Fort Lee, NJ: DAVA Pharmaceuticals, Inc; 2016.
- 11. Neoral (cyclosporine) [package insert]. East Hanover, NJ: Novartis Pharmaceuticals Corporation; 2009.
- 12. Otezla (apremilast) [package insert]. Summit, NJ: Celgene Corporation; 2017.
- 13. Humira (adalimumab) [package insert]. North Chicago, IL: AbbVie Inc; 2017.
- 14. Remicade (infliximab) [package insert]. Horsham, PA: Janssen Biotech, Inc; 2013.
- 15. Stelara (ustekinumab) [package insert]. Horsham, PA: Janssen Biotech, Inc; 2016.
- 16. Cosentyx (sekukinumab) [package insert]. East Hanover, NJ: Novartis Pharmaceuticals Corporation; 2015.
- 17. Taltz (ixekizumab) [package insert]. Indianapolis, IN: Eli Lilly and Company; 2017.

- 18. Siliq (brodalumab) [package insert]. Bridgewater, NJ: Valeant Pharmaceuticals North America LLC; 2017.
- 19. Armstrong AW, Robertson AD, Wu J, et al. Undertreatment, treatment trends, and treatment dissatisfaction among patients with psoriasis and psoriatic arthritis in the United States: findings from the National Psoriasis Foundation surveys, 2003-2011. JAMA Dermatol 2013;149(10):1180-5.
- 20. Papp K, Gordon K, Thaci D, et al. Phase 2 Trial of Selective Tyrosine Kinase 2 Inhibition in Psoriasis. N Engl J Med 2018;379(14):1313-21.
- 21. Watford WT, Hissong BD, Bream JH, et al. Signaling by IL-12 and IL-23 and the immunoregulatory roles of STAT4. Immunol Rev 2004;202:139-56.
- 22. Tokarski JS, Zupa-Fernandez A, Tredup JA, et al. Tyrosine kinase 2-mediated signal transduction in T lymphocytes is blocked by pharmacological stabilization of its pseudokinase domain. J Biol Chem 2015;290(17):11061-74.
- 23. Shaw MH, Boyartchuk V, Wong S, et al. A natural mutation in the Tyk2 pseudokinase domain underlies altered susceptibility of B10.Q/J mice to infection and autoimmunity. Proc Natl Acad Sci U S A 2003;100(20):11594-9.



- 25. Feldman SR, Krueger GG. Psoriasis assessment tools in clinical trials. Ann Rheum Dis 2005;64 Suppl 2:ii65-8; discussion ii9-73.
- 26. Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica 1978;157(4):238-44.





44. Husni ME, Meyer KH, Cohen DS, et al. The PASE questionnaire: pilot-testing a psoriatic arthritis screening and evaluation tool. J Am Acad Dermatol 2007;57(4):581-7.

- 45. Levey AS, Coresh J, Greene T, et al. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med 2006;145(4):247-54.
- 46. Kroenke K, Strine TW, Spitzer RL, et al. The PHQ-8 as a measure of current depression in the general population. J Affect Disord 2009;114(1-3):163-73.
- 47. Dhingra SS, Kroenke K, Zack MM, et al. PHQ-8 Days: a measurement option for DSM-5 Major Depressive Disorder (MDD) severity. Popul Health Metr 2011;9:11.
- 48. Draft Guidance for Industry: Suicidal Ideation and Behavior: Prospective Assessment of Occurrence in Clinical Trials. U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research. Draft August 2012. Publication UCM225130.
- 49. Greist JH, Mundt JC, Gwaltney CJ, et al. Predictive value of baseline electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) assessments for identifying risk of prospective reports of suicidal behavior during research participation. Innov Clin Neurosci 2014;11(9-10):23-31.
- 50. Mundt JC, Greist JH, Jefferson JW, et al. Prediction of suicidal behavior in clinical research by lifetime suicidal ideation and behavior ascertained by the electronic Columbia-Suicide Severity Rating Scale. J Clin Psychiatry 2013;74(9):887-93.
- 51. Posner K, Oquendo MA, Gould M, et al. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry 2007;164(7):1035-43.

| 11 | APPENI | DICES | |
|---|---|---|---|
| APPENDI | X 1 | ABBREVIATIONS AND TRADEMARKS | 83 |
| APPENDI | X 2 | STUDY GOVERNANCE CONSIDERATIONS | 88 |
| APPENDI | X 3 | ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS: DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, FOLLOW-UP AND REPORTING | 96 |
| APPENDI | X 4 | WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND METHODS OF CONTRACEPTION | 100 |
| APPENDI | X 5 | STATIC PHYSICIAN'S GLOBAL ASSESSMENT OF PSORIASIS (sPGA) | 104 |
| APPENDE | X 6 | PSORIASIS AREA AND SEVERITY INDEX (PASI) | 105 |
| APPENDI | X 13 | Classification Criteria for Psoriatic Arthritis (CASPAR) | 113 |
| APPENDI | X 17 | JDA criteria for Severity assessment of pustular psoriasis (generalized psoriasis) | 118 |
| APPENDI | X 23 | PSORIATIC ARTHRITIS SCREENING AND EVALUATION (PASE) QUESTIONNAIRE | 130 |
| APPENDI | X 24 | EIGHT-ITEM PATIENT HEALTH QUESTIONNAIRE (PHQ-8) | 131 |
| APPENDI | X 25 | SUICIDAL IDEATION AND BEHAVIOR CATEGORIES AND DEFINITIONS | 132 |

# APPENDIX 1 ABBREVIATIONS AND TRADEMARKS

| Term Definition | |
|-----------------|-------------------------------------------------|
| ACR | American College of Rheumatology |
| AE | adverse event |
| AEI | Adverse event of interest |
| ALT | alanine aminotransferase |
| Anti-HCV ab | hepatitis C virus antibody |
| AST | aspartate aminotransferase |
| BID | twice daily |
| BMS | Bristol-Myers Squibb |
| BID | twice daily |
| BMS | Bristol-Myers Squibb |
| BP | blood pressure |
| BSA | body surface area |
| BUN | Blood urea nitrogen |
| CASPAR | Classification Criteria for Psoriatic Arthritis |
| CBC | complete blood count |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| CK | creatine phosphokinase |
| CRF | case report form |

| Term | Definition |
|---------|------------------------------------------------------|
| CSR | clinical study report |
| CT | Computed tomography |
| CTA | clinical trial agreement |
| DILI | drug-induced liver injury |
| DLQI | Dermatology Life Quality Index |
| DNA | deoxyribonucleic acid |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| eC-SSRS | electronic Columbia-Suicide Severity Rating<br>Scale |
| eGFR | Estimated Glomerular Filtration Rate |
| EHR | electronic health records |
| EMR | electronic medical records |
| EP | Erythrodermic psoriasis |
| FDA | Food and Drug Administration |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GPP | Generalized pustular psoriasis |
| HBcAb | hepatitis B core antibody |

| Term | Definition |
|-------|-------------------------------------------------------------|
| HbsAb | hepatitis B surface antibody |
| HBsAg | hepatitis B surface antigen |
| HBV | hepatitis B virus |
| hCG | human chorionic gonadotropin |
| Hct | hematocrit |
| HCV | hepatitis C virus |
| HDL | High Density Lipoprotein |
| Hgb | hemoglobin |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HIV | human immunodeficiency virus |
| HRT | hormone replacement therapy |
| IB | Investigator Brochure |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IFN | interferon |
| IgG | immunoglobulin gamma |
| IGRA | interferon gamma release assay |
| IL | interleukin |
| IMP | investigational medicinal product |
| IP | investigational product |
| IRB | Institutional Review Board |
| IRT | interactive response technology |
| IV | intravenous |
| JAK | Janus kinase |
| JDA | Japanese Dermatological Association |
| LAM | lactation amenorrhea method |
| LDH | lactate dehydrogenase |

| Term | Definition |
|-------|----------------------------------------------|
| LDL | low density lipoprotein |
| LTBI | latent tuberculosis infection |
| PASE | psoriatic arthritis screening and evaluation |
| PASI | Psoriasis Area and Severity Index |
| PCR | Polymerase Chain Reaction |
| PD | pharmacodynamics |
| PE | physical examination |
| PCP | phencyclidine |
| PHQ-8 | Eight-Item Patient Health Questionnaire |
| PK | pharmacokinetics |
| PRO | patient reported outcome |
| PsA | psoriatic arthritis |
| PUVA | Psoralens with ultraviolet A |
| QD | once daily |
| QOD | every other day |
| RNA | ribonucleic acid |
| SAE | serious adverse event |
| SIB | Suicidal Ideation and Behavior |

| Term | Definition |
|-------|---------------------------------------------------|
| SOA | schedule of events |
| sPGA | static Physician Global Assessment |
| STAT | signal transducer and activator of transcription |
| SUSAR | Suspected, Unexpected Serious Adverse<br>Reaction |
| T3 | Triiodothyronine |
| T4 | Thyroxine |
| ТВ | tuberculosis |
| TEAE | treatment-emergent adverse event |
| TSH | thyroid-stimulating hormone |
| TNF | tumor necrosis factor |
| TYK2 | tyrosine kinase 2 |
| ULN | upper limit of normal |
| UVB | ultraviolet B |
| WOCBP | women of childbearing potential |
| WHO | World Health Organization |

#### APPENDIX 2 STUDY GOVERNANCE CONSIDERATIONS

## **Regulatory and Ethical Considerations**

### **Good Clinical Practice**

This study will be conducted in accordance with:

- Good Clinical Practice (GCP)
- as defined by the International Council on Harmonisation (ICH)
- in accordance with the ethical principles underlying European Union Directive 2001/20/EC
- United States Code of Federal Regulations, Title 21, Part 50 (21CFR50)
- applicable local requirements.

The study will be conducted in compliance with the protocol. The protocol and any amendments and the subject informed consent will receive approval/favorable opinion by Institutional Review Board/Independent Ethics Committee (IRB/IEC), and regulatory authorities according to applicable local regulations prior to initiation of the study.

All potential serious breaches must be reported to Sponsor or designee immediately. A serious breach is a breach of the conditions and principles of GCP in connection with the study or the protocol, which is likely to affect, to a significant degree, the safety or physical or mental integrity of the subjects of the study or the scientific value of the study.

Personnel involved in conducting this study will be qualified by education, training, and experience to perform their respective tasks.

This study will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (eg, loss of medical licensure, debarment).

## **Institutional Review Board/Independent Ethics Committee**

Before study initiation, the investigator must have written and dated approval/favorable opinion from the IRB/IEC for the protocol, consent form, subject recruitment materials (eg, advertisements), and any other written information to be provided to subjects. The investigator or BMS should also provide the IRB/IEC with a copy of the Investigator Brochure or product labeling information to be provided to subjects and any updates.

The investigator, Sponsor or designee should provide the IRB/IEC with reports, updates and other information (eg, expedited safety reports, amendments, and administrative letters) according to regulatory requirements or institution procedures.

## **Compliance with the Protocol and Protocol Revisions**

The investigator should not implement any deviation or change to the protocol without prior review and documented approval/favorable opinion of an amendment from the IRB/IEC (and if applicable, also by local health authority) except where necessary to eliminate an immediate hazard(s) to study subjects.

If a deviation or change to a protocol is implemented to eliminate an immediate hazard(s) prior to obtaining relevant approval/favorable opinion(s) the deviation or change will be submitted, as soon as possible to:

- IRB/IEC for
- Regulatory Authority(ies), if applicable by local regulations (per national requirements)

Documentation of approval/favorable opinion signed by the chairperson or designee of the IRB(s)/IEC(s) and if applicable, also by local health authority must be sent to BMS.

If an amendment substantially alters the study design or increases the potential risk to the subject: (1) the consent form must be revised and submitted to the IRB(s)/IEC(s) for review and approval/favorable opinion; (2) the revised form must be used to obtain consent from subjects currently enrolled in the study if they are affected by the amendment; and (3) the new form must be used to obtain consent from new subjects prior to enrollment.

If the revision is done via an administrative letter, investigators must inform their IRB(s)/IEC(s).

#### **Financial Disclosure**

Investigators and sub-investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### **Informed Consent Process**

Investigators must ensure that subjects are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which they volunteer to participate.

In situations where consent cannot be given to subjects, their legally acceptable representatives (as per country guidelines) are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which the subject volunteers to participate.

Sponsor or designee will provide the investigator with an appropriate (ie, Global or Local) sample informed consent form which will include all elements required by ICH, GCP, and applicable regulatory requirements. The sample informed consent form will adhere to the ethical principles that have their origin in the Declaration of Helsinki.

## Investigators must:

- Provide a copy of the consent form and written information about the study in the language in which the subject is most proficient prior to clinical study participation. The language must be non-technical and easily understood.
- Allow time necessary for subject or subject's legally acceptable representative to inquire about the details of the study.

- Obtain an informed consent signed and personally dated by the subject or the subject's legally acceptable representative and by the person who conducted the informed consent discussion.
- Obtain the IRB/IEC's written approval/favorable opinion of the written informed consent form and any other information to be provided to the subjects, prior to the beginning of the study, and after any revisions are completed for new information.

If informed consent is initially given by a subject's legally acceptable representative or legal guardian, and the subject subsequently becomes capable of making and communicating his or her informed consent during the study, consent must additionally be obtained from the subject.

Revise the informed consent whenever important new information becomes available that is relevant to the subject's consent. The investigator, or a person designated by the investigator, should fully inform the subject or the subject's legally acceptable representative or legal guardian, of all pertinent aspects of the study and of any new information relevant to the subject's willingness to continue participation in the study. This communication should be documented.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules applicable to regulatory requirements, the subjects' signed ICF and, in the US, the subjects' signed HIPAA Authorization.

The consent form must also include a statement that BMS and regulatory authorities have direct access to subject records.

For minors, according to local legislation, one or both parents or a legally acceptable representative must be informed of the study procedures and must sign the informed consent form approved for the study prior to clinical study participation. The explicit wish of a minor, who is capable of forming an opinion and assessing this information to refuse participation in, or to be withdrawn from, the clinical study at any time should be considered by the investigator.

Minors who are judged to be of an age of reason must also give their written assent.

Subjects unable to give their written consent (eg, stroke or subjects with or severe dementia) may only be enrolled in the study with the consent of a legally acceptable representative. The subject must also be informed about the nature of the study to the extent compatible with his or her understanding, and should this subject become capable, he or she should personally sign and date the consent form as soon as possible. The explicit wish of a subject who is unable to give his or her written consent, but who is capable of forming an opinion and assessing information to refuse participation in, or to be withdrawn from, the clinical study at any time should be considered by the investigator.

The rights, safety, and well-being of the study subjects are the most important considerations and should prevail over interests of science and society.

#### **Source Documents**

The investigator is responsible for ensuring that the source data are accurate, legible, contemporaneous, original, and attributable, whether the data are hand-written on paper or entered electronically. If source data are created (first entered), modified, maintained, archived, retrieved,

or transmitted electronically via computerized systems (and/or any other kind of electronic devices) as part of regulated clinical trial activities, such systems must be compliant with all applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical/health records (EMRs/EHRs), adverse event tracking/reporting, protocol required assessments, and/or drug accountability records).

When paper records from such systems are used in place of electronic format to perform regulated activities, such paper records should be certified copies. A certified copy consists of a copy of original information that has been verified, as indicated by a dated signature, as an exact copy having all of the same attributes and information as the original.

## **Study Treatment Records**

Records for study treatments (whether supplied by BMS, its vendors, or the site) must substantiate study treatment integrity and traceability from receipt, preparation, administration, and through destruction or return. Records must be made available for review at the request of BMS/designee or a health authority.

| If | Then |
|---|---|
| Supplied by BMS (or its vendors): | Records or logs must comply with applicable regulations and guidelines and should include: • amount received and placed in storage area |
| | amount currently in storage area |
| | • label identification number or batch number |
| | • amount dispensed to and returned by each subject, including unique subject identifiers |
| | • amount transferred to another area/site for dispensing or storage |
| | • nonstudy disposition (eg, lost, wasted) |
| | • amount destroyed at study site, if applicable |
| | • amount returned to BMS |
| | • retain samples for bioavailability/bioequivalence, if applicable |
| | • dates and initials of person responsible for Investigational Product |

| If | Then |
|---|---|
| | dispensing/accountability, as per the Delegation of Authority Form. |
| Sourced by site, and not supplied by BMS or its vendors (examples include IP sourced from the sites stock or commercial supply, or a specialty pharmacy) | The investigator or designee accepts responsibility for documenting traceability and study treatment integrity in accordance with requirements applicable under law and the SOPs/standards of the sourcing pharmacy. These records should include: • label identification number or batch number • amount dispensed to and returned by each subject, including unique subject identifiers • dates and initials of person responsible for Investigational Product dispensing/accountability, as per the Delegation of Authority Form. |

BMS or designee will provide forms to facilitate inventory control if the investigational site does not have an established system that meets these requirements.

### **Case Report Forms**

An investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the investigation on each individual treated or entered as a control in the investigation. Data that are derived from source documents and reported on the CRF must be consistent with the source documents or the discrepancies must be explained. Additional clinical information may be collected and analyzed in an effort to enhance understanding of product safety. CRFs may be requested for AEs and/or laboratory abnormalities that are reported or identified during the course of the study.

For sites using the Sponsor or designee electronic data capture tool, electronic CRFs will be prepared for all data collection fields except for fields specific to SAEs and pregnancy, which will be reported on the electronic SAE form and paper Pregnancy Surveillance Form, respectively. If electronic SAE form is not available, a paper SAE form can be used.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules in accordance with the applicable regulatory requirement(s).

The investigator will maintain a signature sheet to document signatures and initials of all persons authorized to make entries and/or corrections on CRFs.

The completed CRF, SAE/pregnancy CRFs, must be promptly reviewed, signed, and dated by the investigator or qualified physician who is a subinvestigator and who is delegated this task on the Delegation of Authority Form. Sub-investigators in Japan may not be delegated the CRF approval task. For electronic CRFs, review and approval/signature is completed electronically through the electronic data capture tool. The investigator must retain a copy of the CRFs including records of the changes and corrections.

Each individual electronically signing electronic CRFs must meet Sponsor or designee training requirements and must only access the electronic data capture tool using the unique user account provided by Sponsor or designee. User accounts are not to be shared or reassigned to other individuals

## **Monitoring**

Sponsor or designee representatives will review data centrally to identify potential issues to determine a schedule of on-site visits for targeted review of study records.

Representatives of BMS must be allowed to visit all study site locations periodically to assess the data quality and study integrity. On site they will review study records and directly compare them with source documents, discuss the conduct of the study with the investigator, and verify that the facilities remain acceptable. Certain CRF pages and/or electronic files may serve as the source documents.

In addition, the study may be evaluated by Sponsor or designee internal auditors and government inspectors who must be allowed access to CRFs, source documents, other study files, and study facilities. BMS audit reports will be kept confidential.

The investigator must notify BMS promptly of any inspections scheduled by regulatory authorities, and promptly forward copies of inspection reports to Sponsor or designee.

#### **Records Retention**

The investigator (or head of the study site in Japan) must retain all study records and source documents for the maximum period required by applicable regulations and guidelines, or institution procedures, or for the period specified by BMS or designee, whichever is longer. The investigator (or head of the study site in Japan) must contact BMS prior to destroying any records associated with the study.

BMS or designee will notify the investigator (or head of the study site in Japan) when the study records are no longer needed.

If the investigator withdraws from the study (eg, relocation, retirement), the records shall be transferred to a mutually agreed upon designee (eg, another investigator, study site, IRB). Notice of such transfer will be given in writing to BMS or designee.

## **Return of Study Treatment**

For this study, study treatments (those supplied by BMS, a vendor or sourced by the investigator) such as partially used study treatment containers, vials and syringes may be destroyed on site.

| If | Then |
|---|---|
| Study treatments supplied by BMS (including its vendors) | Any unused study treatments supplied by BMS can only be destroyed after being inspected and reconciled by the responsible Study Monitor unless study treatments containers must be immediately destroyed as required for safety, or to meet local regulations (eg, cytotoxics or biologics). |
| | If study treatments will be returned, the return will be arranged by the responsible Study Monitor. |
| Study treatments sourced by site, not supplied<br>by BMS (or its vendors) (examples include<br>study treatments sourced from the sites stock<br>or commercial supply, or a specialty<br>pharmacy) | It is the investigator's or designee's responsibility to dispose of all containers according to the institutional guidelines and procedures. |

It is the investigator's or designee's responsibility to arrange for disposal, provided that procedures for proper disposal have been established according to applicable federal, state, local, and institutional guidelines and procedures, and provided that appropriate records of disposal are kept. The following minimal standards must be met:

- On-site disposal practices must not expose humans to risks from the drug.
- On-site disposal practices and procedures are in agreement with applicable laws and regulations, including any special requirements for controlled or hazardous substances.
- Written procedures for on-site disposal are available and followed. The procedures must be filed with the site's SOPs and a copy provided to BMS upon request.
- Records are maintained that allow for traceability of each container, including the date disposed of, quantity disposed, and identification of the person disposing the containers. The method of disposal, ie, incinerator, licensed sanitary landfill, or licensed waste disposal vendor must be documented.
- Accountability and disposal records are complete, up-to-date, and available for the Monitor to review throughout the clinical trial period.

It is the investigator's or designee's responsibility to arrange for disposal of all empty containers.

If conditions for destruction cannot be met the responsible Study Monitor will make arrangements for return of study treatments provided by BMS (or its vendors). Destruction of non-study

treatments sourced by the site, not supplied by BMS, is solely the responsibility of the investigator or designee.

## **Clinical Study Report and Publications**

A Signatory Investigator must be selected to sign the clinical study report.

For this protocol, the Signatory Investigator will be selected as appropriate based on the following criteria:

- External Principal Investigator designated at protocol development
- National Coordinating Investigator
- Study Steering Committee chair or their designee
- Subject recruitment (eg, among the top quartile of enrollers)
- Involvement in trial design
- Regional representation (eg, among top quartile of enrollers from a specified region or country)
- Other criteria (as determined by the study team)

The data collected during this study are confidential and proprietary to Sponsor or designee. Any publications or abstracts arising from this study must adhere to the publication requirements set forth in the clinical trial agreement (CTA) governing study site or investigator participation in the study. These requirements include, but are not limited to, submitting proposed publications to Sponsor or designee at the earliest practicable time prior to submission or presentation and otherwise within the time period set forth in the CTA.

### **APPENDIX 3**

# ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS: DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, FOLLOW-UP AND REPORTING

#### **Adverse Events**

### **Adverse Event Definition:**

An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.

# **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or results from other safety assessments (eg, ECG, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator. Note that abnormal lab tests or other safety assessments should only be reported as AEs if the final diagnosis is not available. Once the final diagnosis is known, the reported term should be updated to be the diagnosis.
- Exacerbation of a chronic or intermittent preexisting condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study
  intervention or a concomitant medication. Overdose, as a verbatim term (as reported by
  the investigator), should not be reported as an AE/SAE unless it is an intentional
  overdose taken with possible suicidal/self-harming intent. Such overdoses should be
  reported regardless of sequelae and should specify "intentional overdose" as the
  verbatim term.

### **Events NOT Meeting the AE Definition**

- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).

# **DEFINITION OF SAE**

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met.

#### SERIOUS ADVERSE EVENTS

## Serious Adverse Event Definition: Any untoward medical occurrence that, at any dose:

Results in death

Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)

Requires inpatient hospitalization or causes prolongation of existing hospitalization (see note below)

Note: The following hospitalizations are not considered SAEs in BMS clinical studies:

- a visit to the emergency room or other hospital department < 24 hours, that does not result in admission (unless considered an important medical or life-threatening event)
- elective surgery, planned prior to signing consent
- admissions as per protocol for a planned medical/surgical procedure
- routine health assessment requiring admission for baseline/trending of health status (eg, routine colonoscopy)
- medical/surgical admission other than to remedy ill health and planned prior to entry into the study. Appropriate documentation is required in these cases.
- admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention (eg, lack of housing, economic inadequacy, caregiver respite, family circumstances, administrative reason)
- admission for administration of anticancer therapy in the absence of any other SAEs (applies to oncology protocols)

Results in persistent or significant disability or permanent damage

Is a congenital anomaly/birth defect

Is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the participant or may require intervention [eg, medical, surgical] to prevent one of the other serious outcomes listed in the definition above). Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization. Potential drug-induced liver injury (DILI) is also considered an important medical event (see Section 8.2.8 for the definition of potential DILI).

Pregnancy and potential DILI must follow the same transmission timing and processes to BMS as used for SAEs (see Section 8.2.5 for reporting pregnancies).

#### **EVALUATING AES AND SAES**

## **Assessment of Intensity**

The intensity of AEs is determined by a physician and will use the following levels:

- Mild: An event that is easily tolerated by the subject, causing minimal discomfort, and not interfering with everyday activities.
- Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event; and both AEs and SAEs can be assessed as severe.

# **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE. A "reasonable possibility of a relationship" conveys that there are facts, evidences, and/or arguments to suggest a causal relationship rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the Investigator's Brochure (IB) and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to Sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to Sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send a SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

# Follow-up of AEs and SAEs

If only limited information is initially available, follow-up reports are required. Note: Follow-up SAE reports must include the same investigator term(s) initially reported.

If an ongoing SAE changes in its intensity or relationship to study drug or if new information becomes available, the SAE report must be updated and submitted within 24 hours to BMS (or designee) using the same procedure used for transmitting the initial SAE report.

All SAEs must be followed to resolution or stabilization.

#### REPORTING OF SAES TO SPONSOR OR DESIGNEE

SAEs, whether related or not related to study drug, and pregnancies must be reported to Drug Safety within 24 hours of awareness of the event.

SAEs must be recorded on the SAE Report Form. For studies capturing SAEs through electronic data capture, electronic submission is the required method for reporting. In the event the electronic system is unavailable for transmission, paper forms must be used and submitted immediately. When paper forms are used, the original paper forms are to remain on site.

Pregnancies must be recorded on a paper Pregnancy Surveillance Form and transmitted via email or confirmed facsimile (fax) transmission to:

# APPENDIX 4 WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND METHODS OF CONTRACEPTION

#### **DEFINITIONS**

## **Woman of Childbearing Potential (WOCBP)**

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

## Women in the following categories are not considered WOCBP

- Premenarchal
- Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of the subject's medical records, medical examination, or medical history interview.

- Postmenopausal female
  - A postmenopausal state is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle-stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.

Note: Females treated with hormone replacement therapy (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The duration of the washout period below are suggested guidelines and the investigators should use their judgment in checking serum FSH levels.

- 1 week minimum for vaginal hormonal products (rings, creams, gels)
- 4 week minimum for transdermal products
- 8 week minimum for oral products

Other parenteral products may require washout periods as long as 6 months. If the serum FSH level is > 40 mIU/ml at any time during the washout period, the woman can be considered postmenopausal.

# CONTRACEPTION GUIDANCE FOR FEMALE SUBJECTS OF CHILD BEARING POTENTIAL

One of the highly effective methods of contraception listed below is required during study duration and until the end of relevant systemic exposure, defined as 3 days after the end of study treatment, plus 30 days.

Local laws and regulations may require use of alternative and/or additional contraception methods.

# **Highly Effective Contraceptive Methods That Are User Dependent**

Failure rate of <1% per year when used consistently and correctly.<sup>a</sup>

- Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation<sup>b</sup>
  - oral
  - intravaginal<sup>d</sup>
  - transdermal<sup>d</sup>
- Progestogen-only hormonal contraception associated with inhibition of ovulation<sup>b</sup>
  - oral
  - injectable<sup>d</sup>

## **Highly Effective Methods That Are User Independent**

- Implantable progestogen-only hormonal contraception associated with inhibition of ovulation<sup>bd</sup>
- Intrauterine device<sup>cd</sup>
- Intrauterine hormone-releasing system<sup>cd</sup>
- Bilateral tubal occlusion
- Vasectomized partner

A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

#### Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the subject.

- It is not necessary to use any other method of contraception when complete abstinence is elected.
- WOCBP subjects who choose complete abstinence must continue to have pregnancy tests, as specified in Section 5.1.
- Acceptable alternate methods of highly effective contraception must be discussed in the event that the WOCBP subjects chooses to forego complete abstinence.

#### NOTES:

- Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for subjects participating in clinical studies.
- Hormonal contraception may be susceptible to interaction with the study treatment, which may reduce the efficacy of the contraceptive method. Hormonal contraception is permissible only when there is sufficient evidence that the IMP and other study medications will not alter hormonal exposures such that contraception would be ineffective or result in increased exposures that could be potentially hazardous. In this case, alternative methods of contraception should be utilized.
- Intrauterine devices and intrauterine hormone-releasing systems are acceptable methods of contraception in the absence of definitive drug interaction studies when hormone exposures from intrauterine devices do not alter contraception effectiveness.
- d These methods are not approved nor certified in Japan.

# Less Than Highly Effective Contraceptive Methods That Are User Dependent

Failure rate of >1% per year when used consistently and correctly.

- Male condom with spermicide<sup>a</sup> or male condom without spermicide or male condom applied spermicide
- Female condom with spermicide<sup>a</sup> or without spermicide<sup>a</sup>
- Diaphragm with spermicide<sup>a</sup>
- Cervical cap with spermicide<sup>a</sup>
- Vaginal Sponge with spermicide<sup>a</sup>

• Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mechanism of action

# **Unacceptable Methods of Contraception**

- Periodic abstinence (calendar, symptothermal, post-ovulation methods)
- Withdrawal(coitus interruptus).
- Spermicide only
- Lactation amenorrhea method (LAM)

# CONTRACEPTION GUIDANCE FOR MALE SUBJECTS WITH PARTNER(S) OF CHILD BEARING POTENTIAL.

Male subjects with female partners of childbearing potential are eligible to participate if they agree to the following during the treatment and until the end of relevant systemic exposure.

- Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator.
- Male subjects are required to use a condom for study duration and until the end of relevant systemic exposure defined as 3 days after the end of treatment in the male subject.
- Female partners of males participating in the study to consider use of effective methods of contraception until the end of relevant systemic exposure, defined as 3 days after the end of treatment in the male subject.
- Male subjects with a pregnant or breastfeeding partner must agree to remain abstinent from penile vaginal intercourse or use a male condom during each episode of penile penetration during the treatment and until 3 days after the end of treatment.
- Refrain from donating sperm for the duration of the study treatment and for 3 days after the end of treatment.

#### COLLECTION OF PREGNANCY INFORMATION

Guidance for collection of Pregnancy Information and outcome of pregnancy on the Pregnancy Surveillance Form is provided in Section 8.2.5 and APPENDIX 3.

# APPENDIX 5 STATIC PHYSICIAN'S GLOBAL ASSESSMENT OF PSORIASIS (sPGA)

The static PGA is used to determine the subject's psoriasis lesions overall at a given time point. Overall lesions will be graded for erythema, induration, and scaling based on the scales below. The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score.

| Characteristics | Score | Rating Score |
|---|---|---|
| Erythema (E) (averaged over the whole body) | | 0 = No evidence of erythema, but post inflammatory hyper/hypopigmentation changes may be present 1 = Faint erythema 2 = Light red coloration 3 = Moderate red coloration 4 = Bright red coloration |
| Induration (I) (averaged over the whole body) | | <ul> <li>0 = No evidence of plaque elevation</li> <li>1 = Minimal plaque elevation, barely palpable, = 0.25 mm</li> <li>2 = Mild plaque elevation, slight but definite elevation, indistinct edge, = 0.5 mm</li> <li>3 = Moderate plaque elevation, elevated with distinct edges, = 0.75 mm</li> <li>4 = Severe plaque elevation, hard/sharp borders, ≥ 1 mm</li> </ul> |
| Scaling (S) (averaged over the whole body) | | 0 = No evidence of scaling 1 = Minimal; occasional fine scaling 2 = Mild; fine scale dominates 3 = Moderate; coarse scale predominates 4 = Severe; thick scale predominates |

E + I + S = /3 = (Total Average)

Physician's Static Global Assessment based upon above Total Average

- 0 = Clear, except for residual discoloration
- 1 = Almost clear -majority of lesions have individual scores for E + I + S / 3 that averages 1
- 2 = Mild -majority of lesions have individual scores for E + I + S / 3 that averages 2
- 3 = Moderate majority of lesions have individual scores for E + I + S / 3 that averages 3
- 4 =Severe -majority of lesions have individual scores for E + I + S / 3 that averages 4

Note: Scores should be rounded to the nearest whole number. If total  $\leq 1.49$ , score = 1; if total  $\geq 1.50$ , score = 2.

# APPENDIX 6 PSORIASIS AREA AND SEVERITY INDEX (PASI)

Psoriasis Area and Severity Index (PASI); a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance. Please complete **all** sections of the table and shade in the affected areas on the body diagrams below.

| | Rating score | Body region (and weighting factor) | | | |
|---|---|---|---|---|---|
| Plaque Characteristic | | Head | Upper Extremities | Trunk | Lower Extremities |
| Erythema (Redness) | 0 = None<br>1 = Slight | | | | |
| Infiltration (Thickness) | 2 = Moderate | | | | |
| Desquamation (Scaling) | 3 = Severe<br>4 = Very severe | | | | |
| Add together each of the | 3 scores for each of | the body regions to g | jive 4 separate sub tot | als. | |
| | Sub Totals | A1 = | A2 = | A3 = | A4 = |
| Multiply each sub total by<br>extremities, A3 x 0.3 for t | | | | | |
| | | A1 x 0.1 = B1 | $A2 \times 0.2 = B2$ | $A3 \times 0.3 = B3$ | $A4 \times 0.4 = B4$ |
| | | B1 = | B2 = | B3 = | B4 = |
| Degree of involvement<br>as % for each body<br>region affected; (score<br>each region with score<br>between 0-6) | 0 = None<br>1 = 1-9 %<br>2 = 10-29%<br>3 = 30-49%<br>4 = 50 -69%<br>5 = 70-89%<br>6 = 90-100% | | | | |
| For each body region multiply sub total B1, B2, B3 and B4 by the score (0-6) of the % of body region involved to give 4 subtotals | | | | | |
| C1, C2, C3 and C4 | | | | | |
| | | B1 x score = C1 | B2 x score = C2 | B3 x score = C3 | B4 x score = C4 |
| | | C1 = | C2 = | C3 = | C4 = |
| The patient's PASI scor | e is the sum of C1 | + C2 + C3 + C4 | | PASI= | |














# APPENDIX 13 CLASSIFICATION CRITERIA FOR PSORIATIC ARTHRITIS (CASPAR)

To meet the CASPAR (Classification criteria for Psoriatic ARthritis) criteria, a subject must have inflammatory articular disease (joint, spine, or entheseal) with 3 points from the following 5 categories:

Current psoriasis is assigned 2 points, while all other features are assigned a score of 1.

- 1. Evidence of current psoriasis, a personal history of psoriasis, or a family history of psoriasis. Current psoriasis is defined as psoriatic skin or scalp disease present today as judged by a rheumatologist or dermatologist. A personal history of psoriasis is defined as a history of psoriasis that may be obtained from a patient, family physician, dermatologist, rheumatologist, or other qualified health care provider. A family history of psoriasis is defined as a history of psoriasis in a first-or second-degree relative according to patient report
- 2. Typical psoriatic nail dystrophy including onycholysis, pitting, and hyperkeratosis observed on current physical examination.
- 3. A negative test result for the presence of rheumatoid factor by any method except latex but preferably by enzyme-linked immunosorbent assay or nephelometry, according to the local laboratory reference range.
- 4. Either current dactylitis, defined as swelling of an entire digit, or a history of dactylitis recorded by a rheumatologist.
- 5. Radiographic evidence of juxtaarticular new bone formation, appearing as ill-defined ossification near joint margins (but excluding osteophyte formation) on plain radiographs of the hand or foot.









# APPENDIX 17 JDA CRITERIA FOR SEVERITY ASSESSMENT OF PUSTULAR PSORIASIS (GENERALIZED PSORIASIS)

| Severity assessment of pustular psoriasis (general | ized psoriasis) | | | |
|---|---|---|---|---|
| A. Evaluation of skin symptoms: | Erythema, cyst, edema (0 to 9) | | | |
| B. Evaluation of systemic symptoms and laboratory findings: | | Pyrexia, WBC count, serum CRP, serum albumin (0 to 8) | | |
| oSeverity scale: | Mild | Mod | Severe | |
| (Total score) | (0 to 6) | (7 to 10) | | (11 to 17) |
| A. Evaluation of skin symptoms (0 to 9) | | | | |
| | Severe | Moderate | Mild | None |
| Area of erythematous lesion (total)* | 3 | 2 | 1 | 0 |
| Area of erythematous lesion with pustula ** | 3 | 2 | 1 | 0 |
| Area of edema lesion** | 3 | 2 | 1 | 0 |
| *Ratio (%) against the body surface area (Severe: | ≥75%, Moderate: | ≥25% and <75%, N | 1ild: <25%) | |
| **Ratio (%) against the body surface area (Severe: ≥50%, Moderate: ≥10% and <50%, Mild: <10%) | | | | |
| B. Evaluation of systemic symptoms and laboratory findings (0 to 8) | | | | |
| Score | 2 | 1 | 1 | |
| Pyrexia (°C) | ≥38.5 | ≥37 and • | ≥37 and <38.5 < | |
| WBC count (/mL) | ≥15,000 | ≥10,000 and <15,000 | | <10,000 |
| CRP (mg/dL) | ≥7.0 | ≥0.3 and | ≥0.3 and <7.0 | |
| Serum albumin (g/dL) | <3.0 | ≥3.0 and | ≥3.0 and <3.8 ≥3.8 | |























# APPENDIX 23 PSORIATIC ARTHRITIS SCREENING AND EVALUATION (PASE) QUESTIONNAIRE

# PSORIATIC ARTHRITIS SCREENING AND EVALUATION (PASE) QUESTIONNAIRE

Please circle or mark <u>ONLY ONE</u> of the five choices on the following 15 questions. The answers to these questions will help us better understand your symptoms. This should take about 5 to 6 minutes to complete. Thank you for your time.

| Symptoms sub-scale | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|
| I feel tired for most of the day | 1 | 2 | 3 | 4 | 5 |
| 2. My joints hurt | 1 | 2 | 3 | 4 | 5 |
| 3. My back hurts | 1 | 2 | 3 | 4 | 5 |
| My joints become swollen | 1 | 2 | 3 | 4 | 5 |
| 5. My joints feel 'hot' | 1 | 2 | 3 | 4 | 5 |
| 6. Occasionally, an entire finger or toe becomes swollen, making it look like a 'sausage' | 1 | 2 | 3 | 4 | 5 |
| 7. I have noticed that the pain in my joints moves from one joint to another, eg my wrist will hurt for a few days then my knee will hurt and so on. | 1 | 2 | 3 | 4 | 5 |
| SYMPTOM SCORE (Max 35) | Add scores for questions 1-7 and write in box A | | | | A. |
| Function sub-scale | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
| 8. I feel that my joint problems have affected my ability to work | 1 | 2 | 3 | 4 | 5 |
| 9. My joint problems have affected my ability to care for myself, eg getting dressed or brushing my teeth | 1 | 2 | 3 | 4 | 5 |
| 10. I have had trouble wearing rings on my fingers or my watch | 1 | 2 | 3 | 4 | 5 |
| 11. I have had trouble getting into or out of a car | 1 | 2 | 3 | 4 | 5 |
| 12. I am unable to be as active as I used to be | 1 | 2 | 3 | 4 | 5 |
| 13. I feel stiff for more than 2 hours after waking up in the morning | 1 | 2 | 3 | 4 | 5 |
| 14. The morning is the worst time of day for me | 1 | 2 | 3 | 4 | 5 |
| 15. It takes me a few minutes to get moving to the best of my ability, any time of the day | 1 | 2 | 3 | 4 | 5 |
| FUNCTION SCORE (Max 40) | Add scores for questions 8-15 and write in box B | | | | B. |
| TOTAL PASE SCORE (Max 75) | Add scores in boxes A and B and write in box C | | | | C. |

### APPENDIX 24 EIGHT-ITEM PATIENT HEALTH QUESTIONNAIRE (PHQ-8)

The eight-item Patient Health Questionnaire depression scale is established as a valid self-administered diagnostic and severity measure for depressive disorders. It consists of 8 different questions, with an answer scale from 0 to 3. The overall score is determined by adding up each of the individual answers from each question.

Scoring interpretation is as follows: 0 to 4 no significant depressive symptoms, 5 to 9 mild depressive symptoms, 10 to 14 moderate depressive symptoms, 15 to 19 moderately severe depressive symptoms, and 20 to 24 severe depressive symptoms

# Over the last 2 weeks, how often have you been bothered by any of the following problems?

| | Not at all | Several<br>days | More than half the days | Nearly<br>every day |
|---|---|---|---|---|
| Little interest or pleasure in doing things | 0 | 1 | 2 | 3 |
| 2. Feeling down, depressed, or hopeless | 0 | 1 | 2 | 3 |
| Trouble falling or staying asleep, or sleeping too much | 0 | 1 | 2 | 3 |
| 4. Feeling tired or having little energy | 0 | 1 | 2 | 3 |
| 5. Poor appetite or over eating | 0 | 1 | 2 | 3 |
| 6. Feeling bad about yourself, or that you are a failure, or have let yourself or your family down | 0 | 1 | 2 | 3 |
| 7. Trouble concentrating on things, such as reading the newspaper, or watching television | 0 | 1 | 2 | 3 |
| 8. Moving or speaking so slowly that other people could have noticed? Or the opposite, being so fidgety or restless that you have been moving around a lot more than usual | 0 | 1 | 2 | 3 |

Total Score:

#### **APPENDIX 25** SUICIDAL IDEATION AND BEHAVIOR CATEGORIES AND **DEFINITIONS**

#### **Suicidal Ideation**

#### Passive suicidal ideation: wish to be dead

Patient has thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up.

### Active suicidal ideation: nonspecific (no method, intent, or plan)

General nonspecific thoughts of wanting to end one's life or commit suicide (eg, "I've thought about killing myself") without general thoughts of ways to kill oneself/associated methods, intent, or plan during the assessment period.

### Active suicidal ideation: method, but no intent or plan

Patient has thoughts of suicide and has thought of at least one method during the assessment period. This situation is different than a specific plan with time, place, or method details worked out (eg, thought of method to kill self but not a specific plan). Includes person who would say, "I thought about taking an overdose but I never made a specific plan as to when, where, or how I would actually do it . . . and I would never go through with it."

### Active suicidal ideation: method and intent, but no plan

Active suicidal thoughts of killing oneself, and patient reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them."

## Active suicidal ideation: method, intent, and plan

Thoughts of killing oneself with details of plan fully or partially worked out and patient has some intent to carry it out (ie, some degree of intent is implicit in the concept of plan).

#### **Suicidal Behavior**

#### Completed suicide

A self-injurious behavior that resulted in fatality and was associated with at least some intent to die as a result of the act. Evidence that the individual intended to kill him- or herself, at least to some degree, can be explicit or inferred from the behavior or circumstance.

#### Suicide attempt

A potentially self-injurious behavior, associated with at least some intent to die as a result of the act. Evidence that the individual intended to kill him- or herself, at least to some degree, can be explicit or inferred from the behavior or circumstance. A suicide attempt may or may not result in actual injury.

### Interrupted suicide attempt

When the person is interrupted (by an outside circumstance) from starting a potentially self-injurious act (if not for that, actual attempt would have occurred).

### Aborted suicide attempt

When person begins to take steps toward making a suicide attempt, but stops before actually engaging in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops before being stopped by something else.

### Preparatory acts toward imminent suicidal behaviors

This category can include anything beyond a verbalization or thought, but it stops short of a suicide attempt, an interrupted suicide attempt, or an aborted suicide attempt. This might include behaviors related to assembling a specific method (eg, buying pills, purchasing a gun) or preparing for one's death by suicide (eg, giving things away, writing a suicide note).

#### **Self-Injurious Behavior Without Suicidal Intent**

Self-injurious behavior associated with no intent to die. The behavior is intended purely for other reasons, either to relieve distress (often referred to as self-mutilation (eg, superficial cuts or scratches, hitting or banging, or burns)) or to effect change in others or the environment.